# Foundation Fighting Blindness (FFB) Consortium

## **Gyrate Atrophy Ocular and Systemic Study**

**Protocol Identifying Number: GYROS** 

**Funded by:** Foundation Fighting Blindness and Conquering Gyrate Atrophy Foundation

Version Number: 1.2 28-Nov-2022

## **Key Roles and Signature Page Gyrate Atrophy Ocular and Systemic Study**

**Protocol Identifying Number: GYROS** 

Version Number: v1.2 28-Nov-2022

| GYROS Protocol Co-Chair | |
|--------------------------------|-----------------------------|
| Name, degree | Mandeep Singh, M.D. |
| Signature/Date | |
| <b>GYROS Protocol Co-Chair</b> | |
| Name, degree | David Valle, M.D. |
| Signature/Date | |
| JCHR GYROS Protocol Dire | ctor (Sponsor) |
| Name, degree | Allison Ayala, MS |
| Signature/Date | |
| FFB Representative (Funder) | |
| Name, degree | Todd Durham, PhD. |
| Signature/Date | |
| Statistician | |
| Name, degree | Maureen Maguire, PhD, FARVO |
| Signature/Date | |

## TABLE OF CONTENTS

| CHAPTER 1: BACKGROUND INFORMATION | 19 |
|---------------------------------------------------|----|
| 1.1 Introduction | 19 |
| 1.1.1 Clinical | 19 |
| 1.1.2 Metabolism | 19 |
| 1.1.3 Molecular | 20 |
| 1.2 Treatment | 20 |
| 1.2.1 Arginine Restricted Diet (ARD) | 20 |
| 1.2.2 Pyridoxine Supplementation | 21 |
| 1.2.3 Creatine Supplementation | 22 |
| 1.2.4 Proline Supplementation | 22 |
| 1.2.5 Lysine Supplementation | 22 |
| 1.3 Rationale | 22 |
| 1.4 Study Objective | 23 |
| 1.5 Potential Risks and Benefits | 23 |
| 1.5.1 Known Potential Risks | 23 |
| 1.5.2 Known Potential Benefits | 24 |
| 1.5.3 Risk Assessment | 24 |
| 1.6 General Considerations | 24 |
| CHAPTER 2: STUDY ENROLLMENT AND SCREENING | 26 |
| 2.1 Participant Recruitment and Enrollment | 26 |
| 2.1.1 Participant Recruitment Goals and Strategy | |
| 2.1.1.1 Target Study Sample Size | 26 |
| 2.1.1.2 Participant Recruitment | 27 |
| 2.1.1.3 Participant Enrollment | 27 |
| 2.2 Informed Consent and Authorization Procedures | 27 |
| 2.3 Screening Visit | 28 |
| 2.3.1 Eligibility Criteria | 28 |
| 2.3.1.1 Participant Inclusion Criteria | 28 |
| 2.3.1.2 Ocular Inclusion Criteria | 29 |
| 2.3.1.3 Participant Exclusion Criteria | 29 |
| 2.3.1.4 Ocular Exclusion Criteria | 29 |
| 2.3.2 Screening Data Collection and Testing | 30 |
| 2.3.3 Initial Screen Failures | |
| 2.4 Genetic Screening Phase | 32 |

| 2.4.1.1 Genetic Screen Failures | 32 |
|--------------------------------------------------------------|----|
| 2.4.1.2 Genetics Committee Review | 32 |
| 2.5 Final Study Cohort Criteria | 32 |
| CHAPTER 3: BASELINE VISIT | 34 |
| 3.1 Baseline Visit | 34 |
| 3.2 Food Record and Blood Sample Collection | 34 |
| 3.3 Baseline Procedures | 35 |
| 3.3.1 Baseline Data Collection and Testing Cohorts 1 & 2 | 35 |
| 3.3.2 Baseline Data Collection and Testing Cohort 3 | 36 |
| CHAPTER 4: FOLLOW-UP VISITS | |
| 4.1 Follow-up Visits | 38 |
| 4.2 Target Timelines | |
| 4.3 Food Record and Blood Sample Collection | 39 |
| 4.4 Follow-up Procedures | 40 |
| 4.4.1 Follow-up Data Collection and Testing Cohorts 1 & 2 | 40 |
| 4.4.2 Follow-up Data Collection and Testing Cohort 3 | 42 |
| 4.4.3 Unscheduled Visits | 43 |
| CHAPTER 5: TESTING PROCEDURES AND QUESTIONNAIRES | |
| 5.1 Study Procedure Requirements | |
| 5.2 Questionnaires | 48 |
| CHAPTER 6: UNANTICIPATED PROBLEM AND ADVERSE EVENT REPORTING | |
| 6.1 Unanticipated Problems | |
| 6.2 Adverse Events | |
| 6.2.1 Definitions | |
| 6.2.2 Reportable Adverse Events | |
| 6.2.3 Relationship of Adverse Event to Study Procedure | |
| 6.2.4 Severity (Intensity) of Adverse Event | |
| 6.2.5 Expectedness | |
| 6.2.6 Coding of Adverse Events | |
| 6.2.7 Outcome of Adverse Event | |
| 6.3 Timing of Event Reporting | 53 |
| CHAPTER 7: MISCELLANEOUS CONSIDERATIONS | |
| 7.1 New or ongoing Medical Conditions and Medications | |
| 7.1.1 Pre-Existing Condition | |
| 7.1.2 Medical Conditions during the study | 54 |

| 7.1.3 Medications | 54 |
|---|---|
| 7.2 Prohibited Medications, Treatments, and Procedures | 54 |
| 7.2.1 Prohibited Medications and Treatment for OAT-Related Retinal | |
| Degeneration | 54 |
| 7.2.2 Intraocular Surgical Procedures | 55 |
| 7.2.3 Treatment for Cystoid Macular Edema (CME) | 55 |
| 7.3 Pregnancy Reporting | 55 |
| 7.4 Participant Compensation | 55 |
| 7.5 Participant Withdrawal | 55 |
| 7.6 Confidentiality | 55 |
| CHAPTER 8: STATISTICAL CONSIDERATIONS | 56 |
| 8.1 Statistical and Analytical | 56 |
| 8.2 Sample Size | 56 |
| 8.2.1 Sample Size Considerations for Evaluating Percent Change from Baseline to four (4) Years – All Outcomes | 56 |
| 8.2.2 Sample Size Considerations for Comparing Percent Change from Baseline to four (4) Years within Subgroups of Interest – All Outcomes | 57 |
| 8.2.3 Sample Size Considerations for Precision of the Estimate of the Correlation Between Structure-based, Function-based, and Metabolic-based Outcomes and of | |
| the Correlation Between Eyes | |
| 8.2.4 Final Sample Size Justification | |
| 8.3 Data Analysis | |
| 8.3.1 Primary Objective Analysis | 61 |
| CHAPTER 9: DATA COLLECTION AND MONITORING | 64 |
| 9.1 Case Report Forms and Other Data Collection | 64 |
| 9.1.1 Central Lab | 64 |
| 9.1.2 Research Lab | 64 |
| 9.1.3 Central Genetics Auditor (CGA) | 64 |
| 9.1.4 Genetics Committee | 64 |
| 9.1.5 The Johns Hopkins Institute for Clinical and Translational Research (ICTR) Research Nutrition | 65 |
| 9.1.6 Reading Centers | |
| 9.2 Study Records Retention | |
| 9.3 Quality Assurance and Monitoring | |
| 9.4 Protocol Deviations | |
| CHAPTER 10: ETHICS/PROTECTION OF HUMAN PARTICIPANTS | 67 |
| 10.1 Ethical Standard | 67 |

| 10.2 Institutional Review Boards | 67 |
|------------------------------------------------|----|
| 10.3 Informed Consent Process | 67 |
| 10.3.1 Consent Procedures and Documentation | 67 |
| 10.3.2 Participant and Data Confidentiality | 67 |
| 10.3.3 Future Use of Stored Specimens and Data | 68 |
| 10.3.4 Future Use of Ocular Images | 68 |
| CHAPTER 11: REFERENCES | 69 |

## **LIST OF ABBREVIATIONS**

| ABBREVIATION | DEFINITION |
|---|---|
| AE | Adverse Event |
| ARD | Arginine Restricted Diet |
| BCVA | Best corrected visual acuity |
| BRVT | Berkeley Rudimentary Vision Test |
| CC | Coordinating Center |
| CFR | Code of Federal Regulations |
| CGA | Central Genetics Auditor |
| CI | Confidence interval |
| CME | Cystoid macular edema |
| EC | Ethics Committee |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| EVA | Electronic Visual Acuity |
| EZ | Ellipsoid Zone |
| FAF | Fundus Autofluorescence |
| FFB | Foundation Fighting Blindness |
| FST | Full-field stimulus threshold |
| GCP | Good Clinical Practice |
| GA | Gyrate Atrophy |
| ICF | Informed consent form |
| ICH | International Committee of Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| IOP | Intraocular Pressure |
| IRB | Institutional Review Board |
| KKI | Kennedy Krieger Institute |
| LLVA | Low Luminance Visual Acuity |
| LPV-FVQ II | L.V. Prasad-Functional Vision Questionnaire |
| MRDQ | Michigan Retinal Degeneration Questionnaire |
| MP | Microperimetry |
| N | Number or sample size |
| OAT | ornithine-δ-aminotransferase |
| OCTA | Optical coherence tomography angiography |
| OD | Right Eye |
| OS | Left Eye |
| OU | Both eyes |
| PI | Principal investigator |
| PRO | Patient reported outcomes |

| ABBREVIATION | DEFINITION |
|--------------|-------------------------------------------------------------|
| PROMIS®-29 | Patient-Reported Outcomes Measurement Information System |
| PSC | Posterior sub-capsular |
| QA | Quality Assurance |
| QC | Quality Control |
| RBM | Risk-Based Monitoring |
| RP | Retinitis pigmentosa |
| RPE | Retinal pigment epithelium |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SD-OCT | Spectral domain optical coherence tomography |
| SP | Static perimetry |
| VA | Visual acuity |
| ViSIO-PRO | Visual Symptom and Impact Outcomes Patient Reported Outcome |
| VF | Visual Field |
| VPA | Valproic Acid |

## PROTOCOL SUMMARY

| ITEM | DESCRIPTION |
|---|---|
| Title | |
| Précis | GYROS: Gyrate Atrophy Ocular and Systemic Study Gyrate atrophy (GA) is a rare inherited chorioretinal degeneration that is associated with hyperornithinemia, an inborn error of metabolism caused by autosomal recessive mutations in the ornithine aminotransferase ( <i>OAT</i> ) gene. GA is characterized by childhood-onset nyctalopia and sharply demarcated areas of chorioretinal atrophy that initially involve the midperipheral fundus. The atrophic areas typically coalesce and enlarge towards the posterior pole in the second and third decades of life, leading to severe visual field constriction and vision loss if left untreated. The current standard care treatment of GA is an arginine restricted diet that is implemented in practice using dietary protein restriction with essential amino acid supplementation. However, dietary treatment is highly burdensome on patients and negatively impacts quality of life such that only about ~20% of patients can comply. Strict adherence to dietary protein restriction (particularly through adolescence), essential amino acid supplementation, and nutritional management of body weight especially during intercurrent illness and pregnancy are among the challenges of treatment. Periods of suboptimal dietary control led to plasma ornithine elevation and progressive chorioretinal degeneration. To facilitate a future interventional gene therapy clinical trial, there is a need to evaluate natural history of and the relationship between potential clinical trial outcome measures. |
| Objectives | are among the challenges of treatment. Periods of suboptimal dietary control led to plasma ornithine elevation and progressive chorioretinal degeneration. To facilitate |

| ITEM | DESCRIPTION | | | |
|---|---|---|---|---|
| | for ornithine levels over four (4) years in individuals with | | | |
| | disease-causing <i>OAT</i> variants. | | | |
| | The expected impact of the <i>OAT</i> gene natural history study is to inform a fut interventional clinical trial design and implementation, including the following | | | |
| | | tient variability of ornithin | _ | one wing. |
| | | measures of progression of | | eserved |
| | | ts reproducibility, sensitivi | ty to change, an | nd |
| | relationship with other | | 11.0 | |
| | 1 | gression of retinal degener<br>t-reported outcome measur | | |
| | measures are most se | | ies, and determ | ille willeli |
| Impact | | me points and duration for | a planned futu | re treatment |
| | trial. | * | Î | |
| | <b>5.</b> Use variability and in calculations. | nter-eye correlation of outc | omes for trial s | sample size |
| | | or the future trial, including | | |
| | | at points for severity of dis | ease most likel | y to benefit |
| | from treatment. 7 Establish study process | edures and workflows for p | ractical impler | mentation of |
| | | edures in a future trial. | ractical impici | ilentation of |
| | Multicenter, longitudinal, pro | | ıdy. Participan | ts will be |
| Study Design | assigned to one (1) of three ( | 3) Vision Cohorts based or | n visual acuity ( | (VA) and |
| Number of Sites | kinetic visual fields (VF). | | | |
| Number of Sites | Approximately 12 Structural Outcomes: | | | |
| | | Test | E aurin un auri | Reading |
| 1 | Key Assessments | Test | Equipment | Center |
| | Primary: Quantitative | Test | Equipment | Center |
| | Primary: Quantitative measures of progression | Fundus | | |
| | Primary: Quantitative | Fundus autofluorescence | Optos | <b>Center</b> Yes |
| | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized | Fundus | | |
| | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* | Fundus autofluorescence | | |
| | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF | Fundus autofluorescence (FAF) Ultra-Widefield Color | Optos | Yes |
| | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* | Fundus<br>autofluorescence<br>(FAF) | | |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical | Optos | Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography | Optos | Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical coherence tomography | Optos Optos Heidelberg Spectralis Digital camera | Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical coherence tomography | Optos Optos Heidelberg Spectralis Digital camera capable of capturing | Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical coherence tomography | Optos Optos Heidelberg Spectralis Digital camera capable of | Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above Ellipsoid zone (EZ) area Presence and type of cataract (posterior | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical coherence tomography (SD-OCT) | Optos Optos Heidelberg Spectralis Digital camera capable of capturing external eye photos Megapixels of | Yes<br>Yes<br>Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above Ellipsoid zone (EZ) area Presence and type of cataract (posterior subcapsular and cortical | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical coherence tomography | Optos Optos Heidelberg Spectralis Digital camera capable of capturing external eye photos Megapixels of >=3MP Magnification | Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above Ellipsoid zone (EZ) area Presence and type of cataract (posterior | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical coherence tomography (SD-OCT) | Optos Optos Heidelberg Spectralis Digital camera capable of capturing external eye photos Megapixels of >=3MP | Yes<br>Yes<br>Yes |
| Outcomes | Primary: Quantitative measures of progression of the area of preserved retina and of the area of lesions in standardized regions* Primary: Use with FAF for assessments noted above Ellipsoid zone (EZ) area Presence and type of cataract (posterior subcapsular and cortical | Fundus autofluorescence (FAF) Ultra-Widefield Color Photography Spectral domain optical coherence tomography (SD-OCT) | Optos Optos Heidelberg Spectralis Digital camera capable of capturing external eye photos Megapixels of >=3MP Magnification of 30-40 degrees | Yes<br>Yes<br>Yes |

| M | DESCRIPTION | | | | |
|---|---|---|---|---|---|
| | Foveal avascular zone (FAZ) area and macular vessel density | OCTA Ancillary test at subsessites | t of | Pre-<br>Approved<br>list | Yes |
| | *Other approaches to grading m **Ocular exam by investigator v cataract. Functional Outcomes: | | | f presence of nu | clear sclero |
| | Key Assessments | Test | E | quipment | Reading<br>Center |
| | Visual field sensitivity<br>measured with<br>quantitative topographic<br>analysis (Hill of Vision) | Static Perimetry | Octo | opus 900 Pro | Yes |
| | Early Treatment of Diabetic Retinopathy Study (ETDRS) best corrected visual acuity (BCVA) letter score | Visual Acuity | Vist<br>(EV | etronic ual Acuity (A) system ETDRS ets | N/A |
| | Low visual acuity test -<br>for participants unable to<br>see ETDRS letters | Low Visual<br>Acuity | Rud<br>Visi | keley<br>limentary<br>ion Test<br>VT) | N/A |
| | ETDRS best corrected low luminance visual acuity letter score | Low Luminance<br>Visual Acuity<br>(LLVA) | Visu<br>(EV | etronic<br>ual Acuity<br>(A) system<br>ETDRS<br>ets | N/A |
| | Mean macular sensitivity | Fundus-Guided<br>Microperimetry | MA | IA | Yes |
| | Full-field retinal sensitivity | Full-field stimulus<br>threshold (FST)<br>testing to blue,<br>white, and red<br>stimuli | Diaş<br>Esp | gnosys | No |
| | Metabolic Outcomes: • Primary: Plasma ornithing panel and evaluated by a • Primary: Blood spot orniacids panel and evaluated • Secondary: Proline, lysim metabolite: creatine and in plasma amino acids panel Patient Reported Outcomes | central lab ithine level; obtained l by a central lab ne, glutamine, glutama its precursor guanidine l and evaluated by a c | by fa<br>ate, an | sting blood sp<br>rginine, and re<br>ate; obtained b | ot test ami |

| ITEM | DESCRIPTION |
|---|---|
| | <ul> <li>Michigan Retinal Degeneration Questionnaire (MRDQ)</li> <li>Visual Symptom and Impact Outcomes Patient Reported Outcome (ViSIO-PRO)</li> <li>Patient-Reported Outcomes Measurement Information System (PROMIS®-29)</li> <li>Adolescents 12-17 years: <ul> <li>Visual Symptom and Impact Outcomes Patient Reported Outcome (ViSIO-PRO)</li> <li>L. V. Prasad-Functional Vision Questionnaire (LVP-FVQ II)</li> </ul> </li> </ul> |
| Risk Factors of<br>Interest | <ul> <li>Body weight and height</li> <li>Assessment of B6 supplements and daily arginine and protein intake, based on patient-reported food record sheet evaluated by central expert dietician review.</li> <li>Biochemical validation of new and rare variants in <i>OAT</i> gene, based on skin biopsy evaluated by a central lab.</li> <li>Key Eligibility Criteria: <ul> <li>The complete list of eligibility criteria is in Chapter 2.3.1 and must be reviewed at the Screening Visit. All eligibility criteria must be met to enroll into the genetic screening phase. A key subset of those eligibility criteria includes the following.</li> </ul> </li> </ul> |
| Population | <ol> <li>Age ≥ 12 years of age</li> <li>Clinical diagnosis of retinal dystrophy</li> <li>Must meet one of the Genetic Screening Criteria: <ul> <li>At least 2 disease-causing variants in the OAT gene which are homozygous or heterozygous in trans, based on a report from a clinically certified lab (or a report from a research lab that has been pre-approved by the study Genetics Committee), OR</li> <li>At least 2 disease-causing variants in the OAT gene with unknown phase, based on a report from a clinically certified lab (or a report from a research lab that has been pre-approved by the study Genetics Committee), AND must meet both of the following phenotype</li> </ul> </li> </ol> |
| | criteria: (1) Classic fundus appearance of gyrate atrophy (based on investigator discretion), AND (2) Elevated ornithine levels >300 μmol/L (documented on any prior lab report). Participants eligible upon initial screening will continue to the genetic screening |
| | phase. Following the genetic screening phase, to be eligible to <b>enroll in the study cohort</b> , the following must be documented: Final Study Cohort Criteria: Must meet one of the Genetic Screening Criteria and have the genetic criteria confirmed by a Central Genetics Auditor (CGA). |
| Sample Size and<br>Recruitment | Sample size rationale is detailed in <b>Chapter 8.2</b> . Recruitment will be tracked with approximate distribution in three (3) Vision Cohorts. A goal of at least forty-five (45) participants will be enrolled, with approximately twenty-five (25) in Vision Cohort 1, fifteen (15) in Vision Cohort 2, and five (5) in Vision Cohort 3. |

| ITEM | DESCRIPTION | | |
|---|---|---|---|
| Phase | Natural History Study | | |
| Vision Cohort | Vision Cohort Definitions All participants will be designated into one of the following Vision Cohorts based on data entered at the Screening Visit. See Section 2.1.1.1 Target Study Sample Size for the detailed definitions. VF diameter ≥10° in VF diameter <10° in | | |
| Groups | | every meridian | any meridian |
| | 20/80 or better | Vision Cohort 1 | Vision Cohort 2 |
| | 20/100-20/400 | Vision Cohort 2 | Vision Cohort 2 |
| | 20/500 or worse | Vision Cohort 3 | Vision Cohort 3 |
| Participant<br>Duration | From the time of screening until the forty-eight (48) month visit: Approximately fifty-one (51) Months. • Screening – Baseline Visit, sixty (60) days • Baseline Visit – forty-eight (48) month Follow-up Visit, forty-eight (48) months. | | |
| Study Duration (planned) | Sixty-one (61) months from first enrollment until last participant visit | | |
| Protocol<br>Overview/<br>Synopsis | <ol> <li>Investigator reviews patient's current genetic report as meeting the Genetic Screening Criteria and any other eligibility criteria that can be evaluated based on medical history.</li> <li>Consent participant according to overseeing Institutional Review Board (IRB)/Ethics Committee (EC) requirements.</li> <li>Obtain ID on study website to <i>enroll into initial screening</i>.</li> <li>Complete a Screening Visit to determine eligibility, Vision Cohort and Genetic Screening Group. Participants meeting criteria to continue will <i>enroll into the genetic screening phase</i>. <ol> <li>See flow chart in next section for details.</li> </ol> </li> <li>Complete genetic screening, including review of genetic reports by CGA. Participants meeting criteria to continue will <i>enroll into the study cohort</i>. <ol> <li>See flow chart in next section for details.</li> </ol> </li> <li>Participants who <i>enroll into the study cohort</i> will return to the clinic within sixty (60) days of the Screening Visit date to start baseline testing, and no later than two (2) weeks after receiving confirmation of meeting <i>final study cohort criteria</i> from the CGA.</li> <li>Participants will return to the clinic at 12, 24, 36 and 48 months from the baseline visit start date for follow-up visits.</li> <li>After the 48-month follow-up visit, participation in the study, for all three (3) Vision Cohorts, will be completed.</li> </ol> | | |

## SCHEMATIC OF STUDY ENROLLMENT



### SCHEMATIC OF GENETIC SCREENING PHASE



#### Final Study Cohort Criteria

- At least 2 disease-causing variants in the OATgene which are homozygous or heterozygous in trans, based on a report from a clinically certified lab (or a report from a research lab that has been preapproved by the study Genetics Committee)
   OR
- At least 2 disease-causing variants in the OAT gene with unknown phase, based on a report from a
  clinically certified lab (or a report from a research lab that has been pre-approved by the study
  Genetics Committee) AND must meet both of the following phenotype criteria
  - (1) Classic fundus appearance of gyrate atrophy (based on investigator discretion) AND
  - (2) Elevated ornithine levels >300 µmol/L (documented on any prior lab report)

At the end of recruitment, all genetic reports of participants enrolled into the natural history study will be evaluated by the Genetics Committee for the following. This analysis will not change eligibility to be enrolled into study cohort.

- · Interpretation of pathogenicity based on American College of Medical Genetics (ACMG) criteria
- Genetic classifications for analyses

## SCHEDULE OF STUDY VISITS AND PROCEDURES: VISION COHORT 1 & VISION COHORT 2

| Visit | Screening | Baseline | 12M | 24M | 36M | 48M |
|---|---|---|---|---|---|---|
| Visit Target Windows | (Up to Day | (Day 0) <sup>b</sup> | Wk | Wk | Wk | Wk |
| | -60) a | | $52 \pm 4^{c}$ | 104± 4° | 156± 4° | 208± 4 <sup>c</sup> |
| Participant-Level Procedures | | | | | | |
| Informed Consent / Eligibility Assessment | X | | | | | |
| Demographics/Screening Medical History (including pre-existing conditions, | X | | | | | |
| symptomology history, patient-reported daily activities, and medications) | Λ | | | | | |
| Determination of Vision Cohort | X | | | | | |
| 3mm punch skin biopsy <sup>i</sup> | | X | | | | |
| Concomitant Medications | X | X | X | X | X | X |
| Adverse Events | | X | X | X | X | X |
| Patient Reported Outcomes (PROMIS-29, MRDQ, ViSIO-PRO, LVP-FVQ II) <sup>h</sup> | | X | | X | | X |
| Ocular Procedures - All testing performed in each eye | | | | | | |
| Complete Ophthalmic Exam <sup>f</sup> | X | | X | X | X | X |
| Intraocular Pressure <sup>g</sup> | X | | X | X | X | X |
| Visual acuity (including refraction, ETDRS, BRVT if needed, LLVA if needed) | X | | X | X | X | X |
| SD-OCT volume scans (Heidelberg Spectralis) | | X | X | X | X | X |
| SD-OCT vertical and horizontal scans (Heidelberg Spectralis) | | X | X | X | X | X |
| Axial Length and Corneal Curvature measurements | | X | | X | | X |
| Fundus Autofluorescence (FAF) (Optos) | | X | X | X | X | X |
| Ultra-Widefield Color Photo (Optos) | | X | X | X | X | X |
| Optical coherence tomography angiography (OCTA) <sup>j</sup> | | X | X | X | X | X |
| Red reflex photo k | | X | X | X | X | X |
| Full-field Stimulus Threshold (Diagnosys Espion) | | X | X | X | X | X |
| Static perimetry (Octopus 900 Pro) | | X <sup>d</sup> | X | X | X | X |
| Fundus guided microperimetry (MAIA) | | X <sup>d</sup> | X | X | X | X |
| Kinetic VF III4e for Vision Cohort definition only | Xe | | | | | |

- a. All Screening Visit testing must be completed on the same day (except for kinetic VF, as noted below).
- b. Baseline Visit date (defined as the start date of all Baseline testing) must be no later than two (2) weeks after receiving confirmation of meeting *final study cohort criteria* from the CGA. All Baseline testing must be completed within <u>ten (10)</u> days of the Baseline Visit date, except PROs as specified.
- c. All Follow up visit testing must be completed on the same day, except PROs as specified.
- **d.** For static perimetry and microperimetry, all Vision Cohort 1 and 2 participants will complete two (2) tests at baseline. The results will be compared according to the *visual field criteria* to determine if a third test is needed.
- **e.** Historical measurement performed within the last eighteen (18) months prior to the Screening Visit. If a historical measurement is not available, then perform the Kinetic VF III4e at the Screening Visit.
- **f.** Ophthalmic exam includes slit-lamp biomicroscopy and indirect ophthalmoscopy. Whenever possible the site should make its best effort to ensure that the exam takes place at approximately the same time of the day at each visit and with the same equipment.
- g. IOP measurements will be taken prior to pupil dilation.
- h. PROs may be completed in person or remotely any time within six (6) months of the Baseline visit or any time within the allowable window of the associated visit window (not required to be the same day as the rest of the visit). Required PROs depend on age, see outcomes grid.
- i. Collected by certified investigator; sent to JHU/KKI Biochemical Genetics Lab.
- j. If site does not have the equipment that would be required for the ancillary study, then participation in this test will be waived, with approval from the Coordinating Center. Site must use a pre-approved equipment for this test.
- **k.** Digital camera capable of capturing external eye photos, Megapixels of >=3MP, Magnification of 30-40 degrees, Digital camera export in PNG, TIF, DICOM or BMP.

## SCHEDULE OF STUDY VISITS AND PROCEDURES: VISION COHORT 3

| Visit | Screening | Baseline | 12M | 24M | 36M | 48M |
|---|---|---|---|---|---|---|
| Visit Target Windows | (Up to Day | (Day 0) <sup>b</sup> | Wk | Wk<br>104± 4° | Wk | Wk |
| | -60) a | | 52 ± 4° | 104± 4° | 156± 4° | 208± 4° |
| Participant-Level Procedures | | | | | | |
| Informed Consent / Eligibility Assessment | X | | | | | |
| Demographics/Screening Medical History (including pre-existing conditions, | X | | | | | |
| symptomology history, patient-reported daily activities, and medications) | Λ | | | | | |
| Determination of Vision Cohort | X | | | | | |
| 3mm punch skin biopsy <sup>h</sup> | | X | | | | |
| Concomitant Medications | X | X | X | X | X | X |
| Adverse Events | | X | X | X | X | X |
| Patient Reported Outcomes (PROMIS-29, MRDQ, ViSIO-PRO, LVP-FVQ II) <sup>g</sup> | | X | | X | | X |
| Ocular Procedures - All testing performed in each eye | | | | | | |
| Complete Ophthalmic Exam <sup>e</sup> | X | | X | X | X | X |
| Intraocular Pressure <sup>f</sup> | X | | X | X | X | X |
| Visual acuity (including refraction, ETDRS, BRVT if needed, LLVA if needed) | X | | X | X | X | X |
| SD-OCT volume scans (Heidelberg Spectralis) | | X | X | X | X | X |
| SD-OCT vertical and horizontal scans (Heidelberg Spectralis) | | X | X | X | X | X |
| Axial Length and Corneal Curvature measurements | | X | | X | | X |
| Fundus Autofluorescence (FAF) (Optos) | | X | X | X | X | X |
| Ultra-Widefield Color Photo (Optos) | | X | X | X | X | X |
| Optical coherence tomography angiography (OCTA)i | | X | X | X | X | X |
| Red reflex photo j | | X | X | X | X | X |
| Full-field Stimulus Threshold (Diagnosys Espion) | | X | X | X | X | X |
| Kinetic VF III4e for Vision Cohort definition only | X <sup>d</sup> | | | | | |

- a. All Screening Visit testing must be completed on the same day (except for kinetic VF, as noted below).
- b. Baseline Visit date (defined as the start date of all Baseline testing) must be no later than two (2) weeks after receiving confirmation of meeting *final study cohort criteria* from the CGA). All Baseline testing must be completed within <u>ten (10)</u> days of the Baseline Visit date, except PROs as specified.
- c. All Follow up visit testing must be completed on the same day, except PROs as specified.
- d. Historical Kinetic VF III4e if available. Kinetic VF III4e <u>does not</u> need to be performed at screening if a historical measurement is not available.
- e. Ophthalmic exam includes slit-lamp biomicroscopy and indirect ophthalmoscopy. Whenever possible the site should make its best effort to ensure that the exam takes place at approximately the same time of the day at each visit and with the same equipment.
- **f.** IOP measurements will be taken prior to pupil dilation.
- g. PROs may be completed in person or remotely any time within six (6) months of the Baseline visit or any time within the allowable window of the associated visit window (not required to be the same day as the rest of the visit). Required PROs depend on age, see outcomes grid.
- h. Collected by certified investigator; sent to JHU/KKI Biochemical Genetics Lab.
- i. If site does not have the equipment that would be required for the ancillary study, then participation in this test will be waived, with approval from the Coordinating Center. Site must use a pre-approved equipment for this test.
- j. Digital camera capable of capturing external eye photos, Megapixels of >=3MP, Magnification of 30-40 degrees, Digital camera export in PNG, TIF, DICOM or BMP.

## FOOD RECORD AND SAMPLE COLLECTION SCHEDULE FOR ALL VISION COHORTS

| | Screening | Baseline | 4M | 8M | 12M | 16M | 20M | 24M | 28M | 32M | 36M | 40M | 44M | 48M |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinical site coordinator contacts participant <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Three-day food record a | | X | X b | X b | X b | X b | X b | X b | X b | X b | X b | X b | X b | X |
| Target Windows for<br>Sample Collection | | | Wk<br>17 ± 4 | Wk<br>34 ± 4 | Wk<br>52 ± 4 | Wk<br>69 ± 4 | Wk<br>86 ± 4 | Wk<br>104 ± 4 | Wk<br>121 ± 4 | Wk<br>138 ± 4 | Wk<br>156 ± 4 | Wk<br>173 ± 4 | Wk<br>190 ± 4 | Wk<br>208 ± 4 |
| Fasting plasma amino<br>acids <sup>c</sup> | X | X (2) | | | X | | | X | | | X | | | X |
| Fasting blood spot amino acids <sup>d</sup> | | X | $X^{d}$ | X <sup>d</sup> | X | X <sup>d</sup> | X <sup>d</sup> | X | X <sup>d</sup> | X <sup>d</sup> | X | X <sup>d</sup> | X <sup>d</sup> | X |
| Request Albumin Lab<br>Records <sup>e</sup> | | X | | | X | | | X | | | X | | | X |
| Body Weight | | X | | | X | | | X | | | X | | | X |
| Height <sup>f</sup> | | X | | | X | | | X | | | X | | | X |

- a. The Pre-Sample Participant Telephone Contact should occur four (4) ten (10) days prior to scheduled sample collection date. Food record should occur for three (3) days leading up to the sample collection date. For at-home samples, the Post-Sample Collection Telephone Call should be completed within one (1) day after the scheduled sample collection date.
- b. The Food Record is only collected if the participant is on an arginine-restricted diet. If the participant is not following an arginine-restricted diet, then the food record will not be recorded and collected. See Section 4.3 Food Record and Blood Sample Collection for more details.
- c. Baseline only: two (2) fasting plasma samples collected on two (2) different days, within ten (10) days of Baseline Visit date.
- d. Participant and/or caretaker administered remotely. Samples will be collected on all participants.
- e. Request the most recent albumin records from the participant's overseeing physician. The albumin labs will be requested only if the participant is on an arginine-restricted diet.
- f. Height will be measured annually in participants less than twenty-one (21) years of age at enrollment, otherwise height will only be collected at the Baseline Visit.

## **Chapter 1: Background Information**

#### 1.1 Introduction

1

2

11

29

- Gyrate atrophy (GA) of the choroid and retina (GA, OMIM 258870) is a rare and slowly 3
- progressive chorioretinal degeneration that leads to severe loss of vision. The prevalence of GA 4
- is thought to be approximately 1 in 1,500,000 live births worldwide, but in certain populations 5
- (e.g., Finns) is as high as 1:50,000 live births. Inherited as an autosomal recessive trait, the 6
- primary defect in GA is deficiency of the mitochondrial matrix enzyme, ornithine-δ-7
- aminotransferase (OAT) resulting from biallelic loss of function mutations in the OAT gene 8
- located at 10q26. OAT deficiency accounts for the hyperornithinemia (plasma levels are ~15-fold 9
- increased over normal) present in all GA children and adults ingesting an unrestricted diet. 10

#### 1.1.1 Clinical

- The early symptoms of GA include myopia and reduced night vision in late childhood. Disease 12
- progression is characterized by progressive visual field constriction, visual acuity loss, and 13
- reduced daytime vision that invariably culminate in functional and legal blindness by mid-14
- adulthood. Visual disability is typically severe and is associated with difficulties in educational, 15
- vocational, mental, and personal aspects of life. Ophthalmologic exam reveals a pathognomonic 16
- pattern of chorioretinal degeneration starting as punctate lesions in the mid-periphery which 17
- gradually enlarge forming sharply demarcated circular areas of atrophy often with 18
- 19 hyperpigmented margins. Within the circular areas, the atrophy involves the photoreceptor cell
- layer, retinal pigment epithelium (RPE), and choroid. The full field electroretinogram (ERG) 20
- amplitudes are typically reduced by the second decade of life. Over the ensuing decades, the 21
- atrophic lesions increase in number and size, coalescing to form scalloped margins and 22
- progressing toward the posterior pole of the eye. Patients can also develop cystoid macular 23
- edema (CME) usually in the third decade or beyond. In all patients, posterior sub-capsular (PSC) 24
- cataracts develop toward the end of the second decade of life. Aside from their ocular phenotype, 25
- GA patients are healthy. Although, they can have abnormal electroencephalograms (EEGs). 26
- However, the frequency of seizures is not increased. Some have mild proximal muscle weakness 27
- that is not of clinical consequence. 28

#### 1.1.2 Metabolism

- OAT is a pyridoxal phosphate (vitamin B6) dependent homohexameric transaminase, which 30
- catalyzes the reversible conversion of ornithine and  $\alpha$ -ketoglutarate to  $\Delta 1$ -pyrroline-5-31
- carboxylate (P5C) and glutamate. Each *OAT* monomer has a pyridoxal phosphate covalently 32
- bound to lysine 292. P5C is in non-enzymatic equilibrium with glutamate semialdehyde (GSA) 33
- and is an intermediate in the synthesis of glutamate and proline. When arginine levels (derived 34
- from the breakdown of dietary or endogenous protein) are adequate, the net flux of the OAT 35
- reaction is in the direction of P5C synthesis<sup>1</sup>. When dietary arginine is inadequate, the net flux 36
- reverses to favor ornithine synthesis. Thus, the *OAT* reaction serves an anapleurotic function for 37
- the urea cycle and serves a necessary function for de novo arginine synthesis. Loss of this 38
- anapleurotic function explains why a few infants with GA present with arginine deficiency and 39
- neonatal hyperammonemia<sup>1</sup>. OAT activity is expressed in many cell types including high levels 40
- in the RPE but is low to undetectable in photoreceptors<sup>2</sup>. Deficiency of *OAT* was shown to be the 41

primary defect in GA by our group in 1977.<sup>3</sup> *OAT* activity in GA patient fibroblasts is < 5% of control values<sup>2</sup>.

#### 1.1.3 Molecular

44

- The *OAT* gene and cDNA were cloned in 1988 and shortly thereafter the first disease producing
- mutation was identified<sup>4-6</sup>. Since then, more than seventy-five (75) disease causing loss of
- function variants have been identified<sup>2,7</sup>. As with other rare autosomal recessive conditions, the
- 48 frequency of certain disease producing variants is enriched in certain populations. For example,
- in Finland where GA is 5- to 10-fold more frequent than in other populations, most patients are
- 50 homozygous for the *OAT* L402P allele reflecting a founder effect in the ancestors of modern-
- day Finns<sup>6</sup>. A few *OAT* disease alleles encode a Vitamin B6 mutant enzyme, most of these are
- missense variants near the B6 binding lysine 292, e.g. A226V<sup>2,8</sup>.
- Interestingly, ornithine levels are increased in a second, rare, autosomal recessive inborn error,
- 54 the Hyperornithinemia- Hyperammonemia-Homocitrullinuria syndrome (HHHS, OMIM
- 55 238970). The plasma ornithine values in these patients range from 200-1020 µM but are
- 56 generally lower than those observed in GA. HHHS patients have episodic hyperammonemia
- often with a degree of intellectual disability and spasticity. More than 100 patients have been
- reported and only one is known to have retinal abnormalities but without the funduscopic change
- characteristic of GA<sup>9</sup>. It has been shown that the primary defect in HHHS is loss of function
- 60 mutations in the SLC25A15 gene which encodes ORC1 (aka ORNT1), the inner mitochondrial
- 61 membrane carrier protein that transports ornithine from the cytosol into the mitochondrial matrix
- 62 in exchange for matrix citrulline plus H+, an essential step for normal functioning of the urea
- 63  $\text{cycle}^{10,11}$ .

64

66

67

68

69

70

71

72

73

74

75 76

78

#### 1.2 Treatment

- Development of treatment of GA has been hampered by several factors:
  - The disorder is quite rare so that almost no centers have adequate numbers of patients to compare the course of treated versus non-treated individuals.
  - The patients come to medical attention at different ages and given the high allelic heterogeneity, often have different *OAT* genotypes.
  - There is currently no pathophysiologic model explaining the unique sensitivity of the retina to this inborn error of ornithine metabolism.
  - The progress of the untreated disease is slow and there are no systemic manifestations of hyperornithinemia. As an example, patients on diet therapy did not notice any acute negative consequences of going off-diet.
  - There is no well-studied cohort of untreated patients available for comparison to a treated group.
- Despite these challenges, several approaches have been recently reviewed<sup>12</sup>.

#### 1.2.1 Arginine Restricted Diet (ARD)

- When the basic defect in GA was identified, it was determined that since ornithine is derived
- from arginine released by the breakdown of dietary or endogenous protein, a diet which

maintains adequate nutrition but in which natural protein was restricted should reduce ornithine 81 accumulation. Due to the severity of the required protein restriction, essential amino acids (EAA) 82 were added to the diet to avoid deficiencies of these amino acids and care was taken to provide 83 adequate calories, minerals, and vitamins 13-16. This approach was shown to reduce ornithine 84 levels to near normal (< 200 µM) and with supervision can be maintained by some patients for 85 years with no ill effects. Ultimately, > 25 patients started this diet; most found compliance 86 difficult and only a few were able to maintain reduce levels of ornithine for greater than five (5) 87 years<sup>17</sup>. Evaluation of the consequences of systemically reduce ornithine levels on the progress 88 of the retinal degeneration was challenging for the reasons described above. However, based on 89 fundus photos, visual acuity measures, and other tests, in patients followed over five (5) years or 90 more it was concluded that reduction of plasma ornithine slowed or even stopped the retinal 91 degeneration<sup>17</sup>. 92

This clinical impression was supported by two additional lines of evidence, one in patients and the other in a mouse model of GA. First, as described above, there is substantial heterogeneity in the rate of progression of GA, which is explained in part by allelic heterogeneity in the OAT mutations causing GA. To confirm this, intra- vs inter-familial variation was compared in the ocular phenotype in six (6) GA sibling pairs and found that the ocular phenotypes of siblings were more similar than those of unrelated GA patients of a similar age. From this observation, it was reasoned that in families with multiple affected siblings, the older could serve as the best control for the younger. In two (2) families, both siblings were placed, one older and one younger, on an ARD at the same time. The severity of the younger sibling to that of the older was compared when the younger reached the age of the older at the time of institution of an ARD. In both families, the retinal phenotype of the younger, who had been on an ARD for 5-7 years by the time they reached the age of diagnosis of the older (untreated at that point) was far less severe. This observation strongly supported the hypothesis that reduction of ornithine accumulation is beneficial<sup>18</sup>. Second, using gene targeting, a knockout mouse model of GA was produced. Post-weaning, homozygous *OAT* null mice had hyperornithinemia to an extent like human GA patients. Their ERG, retinal histology and ultrastructure were normal at two (2) months of age but by age six (6) months these parameters were clearly abnormal and by twelve (12) months of age they had unrecordable ERGs and a severe generalized retinal degeneration <sup>19</sup>. By contrast, GA mice placed on an ARD at two (2) months of age maintained near normal plasma ornithine levels and at twelve (12) months of age had normal ERGs and completely normal retinal histology and ultrastructure<sup>20</sup>. These unambiguous results strongly indicate that systemic correction of ornithine accumulation prevents retinal degeneration in GA. As described above, however, an ARD poses an adherence challenge and only ~20% of patients can comply, and all require careful and repeated evaluation to ensure adequate nutrition.

#### 1.2.2 Pyridoxine Supplementation

For many inherited enzyme deficiencies involving vitamin B6-dependent enzymes (all transaminases, many decarboxylases), a fraction of the patients exhibited some improvement when treated with pyridoxine, vitamin B6, a precursor of pyridoxal phosphate, the active form of the vitamin. Normal pyridoxine intake is  $\sim 1 \text{mg/day}$  while the therapeutic dose ranges from 200 -500 mg/day. This approach is completed initially on all new GA patients, instructing them to maintain their usual diet and defining a response as a > 30% reduction in ornithine levels. Using these criteria, < 10% of patients respond. In those patients for whom skin fibroblasts are available, B6 responsivity in the *OAT* activity assays was also evaluated. The B6 responsive

93

94

95

96

97

98 99

100

101

102

103

104

105

106

107

108

109

110

111

112

113

114

115

116

117

118

119

120

121

122

123

124

patients identified have not exhibited a complete correction of ornithine levels, and for those 126 whose ornithine concentrations on B6 >200  $\mu$ M, a modified ARD was recommended<sup>8</sup>. 127

### 1.2.3 Creatine Supplementation

128

136

143

152

- The first step in the creatine biosynthetic pathway is catalyzed by arginine: glycine 129
- amidinotransferase (AGAT), a cytosolic enzyme that is inhibited by ornithine, one of the 130
- reaction products. For this reason, hyperornithinemic GA patients have less than 10% of normal 131
- levels of plasma creatine and its degradation product, creatinine<sup>21</sup>. However, trials with creatine therapy have not prevented progression of the retinal degeneration<sup>22-24</sup> and patients with inborn 132
- 133
- errors of creatine biosynthesis and similar reductions in creatine do not have retinal 134
- degeneration<sup>24</sup>. These observations have reduced enthusiasm for creatine treatment. 135

#### 1.2.4 Proline Supplementation

- Plasma proline levels are normal in GA, but some studies have indicated that proline is an 137
- important energy source for RPE cells and largely is derived from ornithine in a pathway that 138
- depends on *OAT* activity<sup>2,25</sup>. Proline crosses the blood brain barrier poorly<sup>2</sup> and dietary 139
- supplementation with proline has been tried in GA with no beneficial effect. However, this 140
- approach may be worth additional studies, especially if advances in understanding the 141
- pathophysiology of GA support a role for reduced proline consumption by the RPE. 142

#### 1.2.5 Lysine Supplementation

- Plasma lysine levels are reduced in GA patients with a mean near the lower limit of normal.<sup>2</sup> 144
- This is because ornithine and lysine share a common dibasic amino acid transporter in the kidney 145
- and the high levels of ornithine compete with lysine to increase renal losses of lysine. If lysine 146
- levels could be maintained at high, supra-normal levels it should be possible to increase urinary 147
- losses of ornithine. Evidence from GA mice and GA patients indicates that this approach works 148
- but requires high doses of oral lysine which many (most) patients do not tolerate. Moreover, to 149
- be effective, lysine levels must be maintained at supra-normal levels which could have 150
- detrimental consequences over the long-term. 151

#### 1.3 Rationale

- The treatment for GA that has produced clearly positive results is systemic reduction of ornithine 153
- with an ARD. This diet is challenging and only a small fraction of patients can maintain the diet. 154
- The results, to date, support the hypothesis that ornithine is directly involved in pathophysiology 155
- and that systemic reduction is sufficient for a therapeutic benefit. Pyridoxine supplementation 156
- treatment should be beneficial in those patients who have B6-responsive OAT mutations 157
- regardless of the pathophysiological mechanism and all patients merit a trial with clear criteria 158
- for a beneficial effect (>30% decrease in plasma ornithine on an unrestricted diet). To date, 159
- depending on *OAT* genotype, only a few GA patients respond. There is little or no evidence 160
- supporting the other therapeutic approaches currently. A well-controlled natural history study 161
- would be extremely valuable for future therapeutic trials. 162
- There is limited information from previous natural history studies of patients with GA<sup>12,26</sup>. The 163
- available information is based on cross-sectional data from small numbers of patients, or from 164
- longitudinal studies that are either short term treatment studies or natural history studies with 165
- outcomes based on outdated imaging and visual function methodology<sup>17</sup>. 166

#### 1.4 Study Objective

176

177

186

187

188

189

190

191

192

193

194

195

196

197

198

199

200

201

202

203

204

205

- Natural History Characterize the natural history of ornithine levels and retinal degeneration
- (RD) associated with disease-causing *OAT* variants in the presence of standard care dietary
- treatment regimens over 4 years.
- 171 **Metabolic-Structure-Function Relationships** Explore the relationships between structural
- and functional RD outcome measures and plasma ornithine levels.
- 173 **Identify Rapid Progressors** Explore the relationship of possible risk factors (genotype,
- phenotype, environmental, comorbidities, and standard care dietary regimen) with severity and
- progression of metabolic, functional, structural, and patient-reported outcomes.

#### 1.5 Potential Risks and Benefits

#### 1.5.1 Known Potential Risks

- 178 Most examination procedures are considered part of standard care for retinal degenerations. This
- study will be capturing information about participants that includes identifiable, personal
- information, like date of birth (if permitted by site's regulatory bodies). The study has procedures
- in place to protect that information. However, there is a chance that a loss of that protection
- could occur. This would be a loss of confidentiality. There are special efforts being made to
- ensure that this does not happen.
- 184 The sections below summarize the risks and discomforts that may occur during the period of
- prospective data collection.
  - Risks associated with testing visual acuity (VA), kinetic perimetry (KP), microperimetry (MP), static perimetry (SP), Optos fundus autofluorescence (FAF), Optos Color Photos, red reflectance photos, Optical coherence tomography angiography (OCT-A), and patient reported outcome (PRO) questionnaires may include boredom and frustration. However, no lasting adverse effects are associated with these noninvasive tests
  - Dilating eye drops will be used as part of the ophthalmic examination and before the spectral domain optical coherence tomography (SD-OCT), full-field stimulus threshold (FST), and MP. Dilating eye drops may sting, cause light-sensitivity, or an allergic reaction. There is a small risk of inducing a narrow-angle glaucoma attack from the pupil dilation. However, all participants will have had prior pupil dilation, usually on multiple occasions. Therefore, the risk is extremely small. If glaucoma occurs, treatment is available.
  - Intraocular Pressure (IOP) Examination: In rare instances, the cornea may be scratched during measurement of IOP. An abrasion like this may be painful, but it heals quickly with no lasting effects. If a participant experiences a corneal abrasion, ophthalmic ointment may be administered, and an eye patch or gauze may be placed over the eye.
  - **Venipuncture**: Blood draws can cause common mild reactions including pain, bruising, or redness at the sampling site. Less common reactions include bleeding from the sampling site, formation of a small blood clot or swelling of the vein and surrounding tissues, and fainting. The risk of local infection is less than 1 in 1000.

- Fingerstick Risks: About two (2) drops of blood will be removed by fingerstick for measuring ornithine, amino acid, and arginine. Pain is common at the time of lancing. In about 1 in 10 cases, a small amount of bleeding under the skin will produce a bruise. A small scar may persist for several weeks. The risk of local infection is less than 1 in 1000.
  - **Skin biopsy:** Complications associated with a three (3) mm punch biopsy of the skin include a brief sting when the local anesthetic (numbing medicine) is injected at the biopsy site, the possibility of local bleeding and bruising, pain, infection, allergic reaction to the numbing medicine used in the procedure, or damage to the structures beneath the skin site (such as an artery or a nerve). A small scar may persist for several years.

#### 1.5.2 Known Potential Benefits

Study participants are not expected to benefit directly from participation in this study.

#### 1.5.3 Risk Assessment

210

211

212

213

214

215

217

218

219

220

221

222

223

224

225

226

227

228

229

230

231

232

233

234

235

236

237

238

239

240

241

- The known potential risks above, except for venipuncture, fingerstick collection and skin biopsy, are standard-of-care procedures that do not pose additional risks to participate in the study.
  - The venipuncture is needed to collect plasma samples to monitor the ornithine levels in relation to progression of Gyrate Atrophy.
  - A fingerstick blood spot collection is needed to obtain a blood spot sample. This will determine if this procedure is comparable to the plasma sample collection in evaluating the ornithine levels over time.
  - A skin biopsy is an incisional procedure of the skin. The potential complications include localized bleeding, scarring, bruising, pain, redness, swelling, and damage to nerves and blood vessels. These complications are rare, and when they occur, are mild and selflimiting. This procedure will be used to collect the participant's cells, which are fibroblasts. These cells will be used to measure the activity of the participant's *OAT* enzyme and the response to vitamin B6. The research goal is to understand the impact of OAT mutations on plasma ornithine levels and retinal degeneration. The skin biopsy is necessary to quantify OAT enzyme activity in each participant as it is not possible to derive this information from the blood sample, thus providing direct confirmation on the pathogenicity and functional severity of the mutation in each subject. This information will inform the analysis of the plasma ornithine and retinal degeneration outcome measures for the duration of this trial and will complement the development of dietary guidelines for treatment trials in slowing the progression of Gyrate Atrophy. The cells can be stored frozen indefinitely with participant consent. These cells can be re-cultured to perform additional studies as needed to provide a better understanding of Gyrate Atrophy.

#### 1.6 General Considerations

- The study is being conducted in compliance with the policies described in the study policies
- 243 document, with the ethical principles that have their origin in the Declaration of Helsinki, with
- 244 the protocol described herein, and with the standards of Good Clinical Practice (GCP).

- Employing a prospective longitudinal study design is advantageous because it reflects a
- systematic method of data collection. This study design incorporates several strategies to
- 247 minimize bias, detailed below, using considerations from "Rare Diseases: Natural History
- 248 Studies for Drug Development: Guidance for Industry, Draft Guidance.<sup>27</sup> These are considered
- standard for treatment trials and will enhance the translation of the data from this study to a
- 250 treatment trial.

253

254

255

256

257

258

259

260

- Establishing standardized testing procedures and specific required equipment for all investigators, leading to greater consistency and precision in the information collected.
  - Training and certification of study staff who will perform primary outcome procedures by a Reading Center. The Reading Center will grade test results in a uniform manner independently from study sites.
    - Use of standard, consistent definitions of pre-existing medical conditions, medications and treatments, and adverse events (AEs) across all clinical sites.
    - A consistent schedule of follow-up visits for all participants with established visit time frames.
    - A coordinating center (CC) is responsible for monitoring the conduct of the study to ensure adherence to protocol.
- When feasible, data will be directly collected in electronic case report forms, which will be considered the source data.

## **Chapter 2: Study Enrollment and Screening**

### 2.1 Participant Recruitment and Enrollment

264

265

284

285

286

287

- Enrollment will proceed with the goal of at least forty-five (45) participants completing the trial.
- Approximately fifty (50) individuals may be enrolled in the study to achieve this goal.
- Participants who have signed consent and started the Screening process may be permitted to
- 269 continue into the trial, if eligible, even if the enrollment goal has been reached.
- 270 Study participants will be recruited from approximately twelve (12) clinical sites worldwide. All
- eligible participants will be included without regard to gender, race, or ethnicity. The primary
- 272 recruitment strategy will be from the patients referred from the Investigators. However,
- 273 recruitment materials may be made available at retinal disorder websites upon IRB approval.
- 274 The target population for GYROS will be patients with GA associated with disease-causing
- variants in the *OAT* gene. The male: female distribution of patients with *OAT*-related retinal
- degeneration is expected to be approximately 1:1, therefore both genders will be eligible to
- 277 enroll. Additionally, *OAT*-related retinal degeneration affects patients of all racial and ethnic
- 278 groups, thus enrollment will be conducted without regard to race or ethnicity.
- 279 It is expected that GYROS enrollment will be representative of the population of patients with
- 280 gyrate atrophy associated with disease-causing variants in the *OAT* gene, including those under
- the age of eighteen (18). GA can impact individuals in the first or second decade of life,
- 282 therefore it is important that children are included in this natural history study to characterize the
- 283 natural history of retinal degeneration in patients with gyrate atrophy.

#### 2.1.1 Participant Recruitment Goals and Strategy

#### 2.1.1.1 Target Study Sample Size

Recruitment will be tracked by three (3) vision cohorts defined below. Reference **Chapter 6.1**Sample size for the rationale.

| <b>Vision Cohort 1</b> | Criteria that must be met in the <b>better eye*</b> at the Screening Visit: |
|---|---|
| Approximately | o visual acuity ETDRS letter score of 54 or more (approximate Snellen |
| Twenty-five (25) | equivalent 20/80 or better) and visual field** diameter 10 degrees or |
| participants | more in every meridian of the central field |
| | Criteria that must be met in the <b>better eye*</b> at the Screening Visit: |
| Vision Cohort 2 | o visual acuity ETDRS letter score of 19-53 (approximate Snellen |
| Approximately | equivalent 20/100 - 20/400) |
| Fifteen (15) | <u>OR</u> |
| participants | o visual acuity ETDRS letter score of 54 or more (approximate Snellen |
| participants | equivalent 20/80 or better) and visual field** diameter less than 10 |
| | degrees in any meridian of the central field. |
| <b>Vision Cohort 3</b> | Criteria that must be met in the <b>better eye</b> * at the Screening Visit: |
| Approximately | o visual acuity ETDRS letter score of 18 or less (approximate Snellen |
| Five (5) | equivalent 20/500 or worse). |
| participants | equivalent 20/300 of worse). |

| *Better eye<br>definition | The <b>better eye</b> is defined as the eye with the better Screening Visit ETDRS visual acuity. However, if both eyes have the same visual acuity, which is defined as the same Snellen equivalent, then the determination will be made at investigator discretion. In this scenario, the investigator will consider the eye with better fixation or clearer ocular media to permit highest quality retinal imaging. |
|---|---|
| **Visual Field | The <b>visual field</b> (VF) is defined as the clinically determined <b>kinetic VF III4e</b> performed within the last 18 months prior to the Screening Visit or performed on the day of the Screening Visit. |

288

| | VF diameter ≥10° in | VF diameter <10° in |
|-----------------|---------------------|---------------------|
| | every meridian | any meridian |
| 20/80 or better | Vision Cohort 1 | Vision Cohort 2 |
| 20/100-20/400 | Vision Cohort 2 | Vision Cohort 2 |
| 20/500 or worse | Vision Cohort 3 | Vision Cohort 3 |

289

290

291

#### 2.1.1.2 Participant Recruitment

The Foundation Fighting Blindness (FFB) Consortium Executive Committee will review recruitment progress and feasibility at regular intervals.

292 293 294

295

296

297

298

Initial recruitment goals will include forty-five (45) participants enrolled into the study vision **cohorts** 1, 2, and 3 combined. If recruitment is not at a rate to meet the initial goals, an interim assessment of feasibility may be made by the FFB Consortium Executive Committee. A minimum of forty (40) participants enrolled in Vision Cohorts 1 and 2 combined will be targeted.

#### 2.1.1.3 Participant Enrollment

299 300 301

and Genetic Screening have been confirmed. This means that potentially more participants will be screened. The number and reasons for screen failures will be tracked. It is possible that

Participants will not be counted as enrolled into the study cohort until Initial Screening

302 303

participants will have completed the screening visit and will be awaiting genetic confirmation at the time the enrolled numbers reach the goals above. Therefore, the final enrolled numbers may

be larger. To limit over-enrollment, clinical sites will be notified as the recruitment goals near 304 completion and efforts will be made to accurately predict numbers in the genetic screening 305

306 queue.

#### 2.2 Informed Consent and Authorization Procedures

308

307

Study participants must be age of majority to consent for themselves, e.g., at least eighteen (18)

years of age in the US. For potential participants who are minors, e.g., under eighteen (18) years 309

of age in the US, a parent/legal guardian (referred to subsequently as "parent") will be provided 310

with the Informed Consent Form to read and will be given the opportunity to ask questions. 311

Potential participants meeting the IRB's minimum age of assent will be given an Assent Form to 312

read and discuss with their parents and study personnel. If the parents and child agree 313

| <ul><li>314</li><li>315</li><li>316</li></ul> | to participate, the Informed Consent Form and Child Assent Form will be signed. A copy of the consent form will be provided to the participant and their parents, and another copy will be added to the participant's study record. |
|---|---|
| 317<br>318<br>319<br>320 | The study protocol will be discussed with the potential study participant by study staff. The potential study participant will be given the Informed Consent Form to read. Potential study participants will be encouraged to discuss the study with family members and their personal physician(s) before deciding whether to participate in the study. |
| 321<br>322<br>323<br>324<br>325 | As part of the informed consent process, each participant will be asked to sign an authorization for release of personal information. The investigator, or his or her designee, will review the study-specific information that will be collected and to whom that information will be disclosed After speaking with the participant, questions will be answered about the details regarding authorization. |
| 326<br>327 | A participant is considered <b>enrolled into the initial screening</b> when the ICF has been signed and a participant ID has been obtained on the study website. |
| 328<br>329 | Participants who become age of majority, e.g., eighteen (18) years of age in the US, during the study will need to re-consent with an adult Informed Consent Form. |
| 330 | 2.3 Screening Visit |
| 331<br>332<br>333<br>334 | After the ICF has been signed, a potential participant will be evaluated for study eligibility through the elicitation of a medical history, performance of ophthalmic tests as described below, and genetic testing, if applicable. The Screening Visit date will be the date the Screening Visit testing procedures started. All Screening Visit testing procedures will be completed on this date. |
| 335 | 2.3.1 Eligibility Criteria |
| 336<br>337 | To be eligible to <b>enroll into the genetic screening phase</b> , a study participant must meet all the inclusion criteria and none of the exclusion criteria at the Screening Visit. |
| 338 | 2.3.1.1 Participant Inclusion Criteria |
| 339<br>340 | Participants must meet all the following inclusion criteria at the Screening Visit to be eligible to enroll into the genetic screening phase. |
| 341<br>342<br>343<br>344<br>345 | <ol> <li>Willing to participate in the study and able to communicate consent during the consent process.</li> <li>Willing and able to complete all study visit assessments at each visit over the forty-eight (48) month study period.</li> <li>Age ≥ 12 years</li> </ol> |
| 346<br>347 | <ul> <li>4. Adult participants must have the capacity to consent on their own behalf.</li> <li>5. Must meet one (1) of the Genetic Screening Criteria below:</li> </ul> |
| 348<br>349<br>350<br>351 | • At least 2 disease-causing variants in the <i>OAT</i> gene which are homozygous or heterozygous in trans, based on a report from a clinically certified lab, or a report from a research lab that has been preapproved by the study Genetics Committee. |
| 352<br>353 | OR |

| 354 | |
|---|---|
| 355 | <ul> <li>At least 2 disease-causing variants in the OAT gene with unknown</li> </ul> |
| 356 | phase, based on a report from a clinically certified lab, or a report from a |
| 357 | research lab that has been pre-approved by the study Genetics Committee, |
| 358 | AND must meet both of the following phenotype criteria: |
| 359 | 1. Classic fundus appearance of gyrate atrophy (based on |
| 360 | investigator discretion) AND |
| 361<br>362 | 2. Elevated ornithine levels >300 μmol/L (documented on any prior lab report). |
| 363 | 2.3.1.2 Ocular Inclusion Criteria |
| 364<br>365 | Participant must meet the following criteria at the Screening Visit to <b>enroll into the genetic screening phase</b> . |
| 366 | <b>6.</b> Both eyes must have a clinical diagnosis of retinal dystrophy |
| 367 | 7. Both eyes must permit good quality photographic imaging (for example, but not |
| 368 | limited to, clear ocular media, adequate pupil dilation, stable fixation). |
| 369 | 2.3.1.3 Participant Exclusion Criteria |
| 370 | Participants must not meet any of the following exclusion criteria at the Screening Visit to be |
| 371 | eligible to enroll into the genetic screening phase. |
| 372 | 1. Single pathogenic or likely pathogenic genetic variants known to be associated with |
| 373 | autosomal dominant retinitis pigmentosa/retinal dystrophy (AD, heterozygous), X- |
| 374 | linked retinitis pigmentosa/retinal dystrophy (XL, hemizygous), or mitochondrial |
| 375 | inheritance. |
| 376 | 2. Expected to enter experimental treatment trial at any time during this study. |
| 377 | 3. History of more than one (1) year of cumulative treatment, at any time, with an agent |
| <ul><li>378</li><li>379</li></ul> | associated with pigmentary retinopathy, including amiodarone, chloroquine, deferoxamine, hydroxychloroquine, pentosan polysulfate, tamoxifen, and |
| 380 | deferoxamine. |
| 381 | Note: Since this is a Natural History Study collecting data on the progression of GA, pregnant |
| 382 | women will not be specifically excluded from participation. |
| 383 | 2.3.1.4 Ocular Exclusion Criteria |
| 384 | If either eye has any of the following ocular exclusion criteria at the Screening Visit, then the |
| 385 | participant is not eligible to enroll into the genetic screening phase. |
| 386 | 4. Current vitreous hemorrhage. |
| 387 | 5. Current complications of pathological myopia (for example, but not limited to, |
| 388 | myopic maculopathy including atrophy, scar, choroidal neovascularization, schisis) |
| 389 | that could inhibit imaging studies of gyrate atrophy-related chorioretinal degeneration |
| 390 | or assessment of visual function. 6. History of introcular surgery (for example, but not limited to cataract surgery) |
| 391 | <b>6.</b> History of intraocular surgery (for example, but not limited to cataract surgery, |

vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months.

- 7. Current or any history of confirmed diagnosis of glaucoma (for example, but not 393 limited to glaucomatous VF changes or nerve changes, or history of glaucoma 394 filtering surgery). 395 **8.** Current or any history of retinal vascular occlusion or proliferative diabetic 396 retinopathy. 397 9. Any clinically significant cystoid macular edema, as determined by the Investigator, 398 that is not stable three (3) months before screening; use of chronic, prophylactic 399 treatment with topical or oral agents (for example, but not limited to, dorzolamide) is 400 allowed. 401 10. History or current evidence of ocular disease that, in the opinion of the investigator, 402 may confound assessment of visual function (for example, but not limited to, 403 tractional or rhegmatogenous retinal detachment, any vitreoretinal surgery, retinal 404 vascular occlusion, proliferative diabetic retinopathy). 405 11. The following medications and treatments are prohibited as they can affect 406 progression of retinitis pigmentosa or confound the assessments. The participant must 407 not have received or plan to receive the following treatments. 408 i. Any use of ocular stem cell or gene therapy: 409 ii. Any treatment with ocriplasmin. 410 iii. Treatment with Ozurdex (dexamethasone), Iluvien or Yutiq (fluocinolone 411 acetonide) intravitreal implant. 412 12. The following medications and treatments are excluded within the specified 413 timeframe: 414 i. Treatment with an ophthalmic oligonucleotide within the last 9 months (last 415 treatment date is less than 9 months prior to Screening Visit date). 416 ii. Treatment with any other product for retinal dystrophy within five times the 417 expected half-life of the product (time from last treatment date to Screening 418 Visit date is at least 5 times the half-life of the given product). 419 iii. Treatment that can alter VA between Screening and Baseline (e.g., 420 periorbital injections. 421 2.3.2 Screening Data Collection and Testing 422 Please reference the schematic of study design at the beginning of the protocol for the flow of the 423 study visit procedures. The following procedures will be performed at the Screening Visit. The 424 testing procedures are detailed in the GYROS Clinical Site Manual of Procedures. An 425 overview of the equipment and technician requirements for all testing is in Chapter 5.1 Study 426 Procedure Requirements. All ocular testing will be performed in each eye, right eye (OD) first 427 and then left eye (OS). Screening procedures will last approximately four (4) hours. 428 429 Participants meeting criteria to continue will be enrolled into the genetic screening phase. 430 Otherwise, the participant will be an initial screen failure. 431
- 432
- The following procedures will be performed, data collected, eligibility criteria checked, and documented at the Screening Visit.
  - 1. Inclusion and exclusion criteria assessed
- 2. Demographics: date of birth, sex, race, and ethnicity

3. Contact information: this will be retained at the site and not entered on the study database 437 4. Medical history: will be elicited from the study participant and extracted from available 438 medical records, including patient-reported daily activities, pre-existing medical 439 conditions, and medications. 440 • Participant will sign a release of medical information form to collect medical 441 records and laboratory records. 442 5. Concomitant medications 443 **6.** Genetic screening assessment, including number and phase of mutations in the *OAT* gene, 444 history of consanguinity, and collection of the source genetic report(s) available at the 445 clinical site. 446 This includes an assessment that the participant meets one of the Genetic 447 Screening Criteria. If the participant does not meet the criteria for one of the 448 Genetic Screening Criteria, then the remainder of procedures and testing are not 449 required. The participant will be discontinued as an **initial screen failure**. 450 7. Complete ophthalmic examination to include: 451 Slit lamp biomicroscopy 452 Indirect ophthalmoscopy 453 **8.** IOP 454 IOP measurements will be taken prior to pupil dilation. 455 9. VA (including refraction, ETDRS, BRVT if needed, LLVA if needed). 456 The VA letter score will determine whether LLVA or BRVT will be performed. 457 The criteria are defined in the GYROS Clinical Site Manual of Procedures. 458 10. Kinetic VF III4e 459 • Vision Cohort 1 and 2: Historical measurement performed within the last 460 eighteen (18) months prior to the Screening Visit. If a historical measurement is 461 not available, then perform the Kinetic VF III4e at the Screening Visit. 462 • Vision Cohort 3: Collect the most recent historical measurement prior to the 463 Screening Visit, if available. Kinetic VF III4e does not need to be performed at 464 screening if a historical measurement is not available. 465 11. Determination of Vision Cohort 466 If the participant's determined Vision Cohort is closed for enrollment, the 467 remainder of procedures and testing are not required. Participant will be 468 discontinued as an initial screen failure. 469

• The Site Personnel will collect one (1) fasting plasma sample.

12. Sample Collection

470

#### 2.3.3 Initial Screen Failures 472 Participants who do not meet criteria to continue as noted above will be discontinued as an 473 initial screen failure. The Screening Visit Form will still be completed, entering "Not Done" for 474 testing not finished. A Final Status Form will be completed, and the reason for screen failure will 475 be noted. 476 2.4 Genetic Screening Phase 477 Participants passing the initial screening and enrolling into the Genetic Screening Phase will 478 submit their genetic lab reports for CGA review. The schematic of study design at the beginning 479 of the protocol summarizes the flow of the Genetic Screening Phase. Reference the GYROS 480 Clinical Site Manual of Procedures for detailed procedures. 481 All genetic reports will be uploaded to the FFB study website by the clinical site. These reports 482 may be reviewed by the CC, associated clinical site, Central Genetics Auditor (CGA), Genetics 483 Committee, and investigators involved in the oversight of the study (which includes the study 484 chair, Operations Committee, and Executive Committee). All genetic reports will be de-485 identified and redacted of all personal data prior to uploading on the FFB study website. 486 The clinical site will upload supporting genetic documentation, including the genetic reports, on 487 the FFB study website. The CGA will review the genetic documentation provided by the clinical 488 site to verify the genetic screening data entry and appropriate documentation of the Genetic 489 Screening Criteria. Additional documentation may be requested as needed to verify the Genetic 490 Screening Criteria and all genetic screening assessments. 491 • If Genetic Screening Criteria are verified, then the participant will be considered 492 enrolled into the study cohort. 493 494 • If the final study cohort is not verified, then the participant will be a genetic screen failure. 495 2.4.1.1 Genetic Screen Failures 496 Participants who do not meet criteria to continue in the study will be discontinued as a genetic 497 screen failure. A Final Status Form will be completed, and the reason for screen failure will be 498 indicated. 499 500 2.4.1.2 Genetics Committee Review A Genetics Committee will review the genetic documentation of participants with verified **final** 501 study cohort criteria and enrolled into the study cohort for interpretation and evaluation of 502

A Genetics Committee will review the genetic documentation of participants with verified **final**study cohort criteria and enrolled into the study cohort for interpretation and evaluation of
whether the *OAT* mutations are causative of the disease (i.e., pathogenic, likely pathogenic).
Cases that are not confirmed as disease causing will remain in the study and will not be
considered ineligible. However, their data may be analyzed separately from those with

506 pathogenic mutations.

507

#### 2.5 Final Study Cohort Criteria

The Final Study Cohort Criteria is participants that meet one of the Genetic Screening

Criteria, and have the genetic criteria confirmed by a Central Genetics Auditor (CGA).

- Participants that meet the initial screening and eligibility criteria, who complete the Genetic
- Screening Phase, and who meet the **final study cohort criteria** will be considered **enrolled into**
- the study cohort. These participants should complete the natural history study.

| 514 | Chapter 3: Baseline Visit |
|---|---|
| 515 | 3.1 Baseline Visit |
| 516<br>517<br>518<br>519 | Participants meeting criteria to enter the natural history study will return for a Baseline Visit within sixty (60) days after receiving confirmation of meeting <b>final study cohort criteria</b> from the CGA. |
| <ul><li>520</li><li>521</li><li>522</li></ul> | The Baseline Visit date will be documented as the date testing procedures began. All Baseline Visit testing procedures will be completed within <u>ten (10) days</u> of the Baseline Visit date, unless specified below. |
| 523 | 3.2 Food Record and Blood Sample Collection |
| 524 | All participants will complete the food record and blood sample collection as described below. |
| 525 | (1) Participant Contact |
| <ul><li>526</li><li>527</li><li>528</li><li>529</li></ul> | The Clinical Site Coordinator will contact the participants (via phone or other remote interface) four (4) to ten (10) days prior to the first of the two (2) scheduled sample collection date. The Pre-Sample Collection Telephone Call will include instructions and reminders of: |
| 530 | o The two (2) sample collection dates. |
| 531 | o Fasting instructions. |
| 532 | <ul> <li>Food record collection instructions.</li> </ul> |
| 533 | (2) Food Record |
| 534<br>535 | The participant will complete a food record to document their daily<br>consumption during the following period: |
| 536 | o <u>Begin</u> three (3) days prior to the first sample collection date |
| 537 | o <u>End</u> one (1) day prior to the last sample collection date |
| <ul><li>538</li><li>539</li><li>540</li></ul> | The participant will digitally send (e-mail or text) a picture of the food record<br>documentation and either mail the original food tracking record to the site or<br>bring it to the site at their Baseline Visit. |
| 541<br>542 | <ul> <li>The Clinical Site Coordinator will enter the data from the food record on the<br/>FFB Study Website.</li> </ul> |
| <ul><li>543</li><li>544</li><li>545</li></ul> | <ul> <li>A Central Dietitian Reviewer (CDR) will review food record on FFB Study<br/>Website to determine nutritional content. This information will be<br/>documented on the FFB Study Website.</li> </ul> |
| 546 | (3) Sample Collection |
| 547 | Site Personnel will collect the following: |
| 548<br>549 | <ul> <li>Two (2) <u>fasting plasma samples</u> on two (2) different days, within ten<br/>(10) days of the Baseline Visit date.</li> </ul> |

| 550<br>551 | | <ul> <li>One (1) <u>fasting blood spot fingerstick</u> on the same day as one of the<br/>fasting plasma samples.</li> </ul> |
|---|---|---|
| <ul><li>552</li><li>553</li></ul> | | <ul> <li>All samples will be shipped to the Kennedy Krieger Institute<br/>(KKI).</li> </ul> |
| <ul><li>554</li><li>555</li><li>556</li></ul> | | The Clinical Site Coordinator would request the most recent lab records with<br>an albumin result if the participant indicated they are currently on an arginine-<br>restricted diet. |
| 557 | 3.3 Baseli | ne Procedures |
| 558<br>559<br>560<br>561<br>562<br>563 | detailed in and certific Requirem | ving procedures will be performed at the Baseline Visit. The testing procedures are a the <b>GYROS</b> Clinical Site Manual of Procedures. An overview of the equipment cation requirements for all testing is in Chapter 5.1: Study Procedure tents. All ocular testing will be performed in each eye, OD first and then OS. Baseline is will last approximately seven (7) – eight (8) hours. Baseline procedures will span 10) days. |
| 564 | 3.3.1 1 | Baseline Data Collection and Testing Cohorts 1 & 2 |
| 565 | 1. | Medical updates to include: |
| 566 | | • New or changed adverse events (AEs) |
| 567 | | <ul> <li>New ocular procedures</li> </ul> |
| 568 | | <ul> <li>New or changed medications</li> </ul> |
| 569 | | <ul> <li>Request medical records and laboratory records if applicable.</li> </ul> |
| 570 | 2. | Patient Reported Outcomes |
| 571 | | ♦ Adults: PROMIS®-29, MRDQ, ViSIO-PRO |
| 572 | | ♦ Adolescents: LPV-FVQ II, ViSIO-PRO |
| 573 | | Children: LPV-FVQ II |
| <ul><li>574</li><li>575</li><li>576</li></ul> | | • The PROs may be completed in person or remotely (phone or other remote methods) any time within six (6) months of the Baseline Visit (not required to be the same day as the rest of the Baseline Visit). |
| 577 | 3. | Skin biopsy (3mm punch skin biopsy) |
| 578 | | • Ship to Johns Hopkins University Department of Genetic Medicine Research Lab |
| 579 | 4. | Spectral Domain Optical Coherence Tomography (SD-OCT) |
| 580 | | Volume Scan |
| 581 | | Vertical and Horizontal Scan |
| 582 | 5. | Axial Length and Corneal Curvature Measurements |
| 583 | 6. | Fundus Autofluorescence |
| 584 | 7. | Widefield color photo |

| 585 | 8. Optical coherence tomography angiography (OCTA) |
|---|---|
| 586 | <ul> <li>Ancillary test; may be waived with approval from the Coordinating Center</li> </ul> |
| 587 | 9. Red reflex photo |
| 588 | 10. Full field Stimulus Threshold (FST) |
| 589 | 11. Static perimetry |
| 590<br>591 | • Two (2) tests will be performed. The clinical site will compare the certified technician determined mean sensitivity from test one (1) versus test two (2). |
| 592<br>593<br>594<br>595 | (a) If the absolute value of the difference between the two tests is ≤ 2.4 dB, then the participant passes static perimetry reliability criteria. A third test is <u>not needed</u> . |
| 596<br>597<br>598 | (b) If the absolute value of the difference between the two tests is > 2.4 dB, then the participant does not pass static perimetry reliability criteria. A third test will be required. |
| 599 | 12. Fundus guided microperimetry |
| 600<br>601 | • Two (2) tests will be performed. The clinical site will compare the certified technician determined mean sensitivity from test one (1) versus test two (2). |
| 602<br>603<br>604<br>605 | (a) If the absolute value of the difference between the two tests divided by the average between them is $\leq 50\%$ OR the absolute value of the difference between the two tests is $\leq 0.5$ dB, then the participant passes the microperimetry reliability criteria. A third test is <u>not needed</u> . |
| 606<br>607<br>608<br>609<br>610 | <b>(b)</b> If the absolute value of the difference between the two tests divided by the average between them is > 50% AND the absolute value of the difference between the two tests is > 0.5 dB, then the participant does not pass microperimetry reliability criteria. A third test will be required. |
| 611 | 13. Measurements to include: |
| 612 | • Weight |
| 613 | • Height |
| 614 | 3.3.2 Baseline Data Collection and Testing Cohort 3 |
| 615 | 1. Medical updates to include |
| 616 | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 617 | <ul> <li>New ocular procedures</li> </ul> |
| | • |
| 618 | New or changed medications |
| 619 | <ul> <li>Request medical records and laboratory records if applicable.</li> </ul> |
| 620 | 2. Patient Reported Outcomes |
| 621 | ◆ Adults: PROMIS®-29, MRDQ, ViSIO-PRO |
| 622 | <ul> <li>Adolescents: LPV-FVQ II, ViSIO-PRO</li> </ul> |
|---|---|
| 623 | • Children: LPV-FVQ II |
| 624<br>625<br>626 | • The PROs may be completed in person or remotely (phone or other remote methods) any time within six (6) months of the Baseline Visit (not required to be the same day as the rest of the Baseline Visit). |
| 627 | 3. Skin biopsy (3mm punch skin biopsy) |
| 628 | • Ship to Johns Hopkins University Department of Genetic Medicine Research Lab |
| 629 | 4. Spectral Domain Optical Coherence Tomography (SD-OCT) |
| 630 | <ul> <li>Volume Scan</li> </ul> |
| 631 | <ul> <li>Vertical and Horizontal Scan</li> </ul> |
| 632 | 5. Axial Length and Corneal Curvature Measurements |
| 633 | 6. Fundus Autofluorescence |
| 634 | 7. Widefield color photo |
| 635 | 8. Optical coherence tomography angiography (OCTA) |
| 636 | <ul> <li>Ancillary test; may be waived with approval from the Coordinating Center</li> </ul> |
| 637 | 9. Red reflex photo |
| 638 | 10. Full field Stimulus Threshold (FST) |
| 639 | 11. Measurements to include: |
| 640 | • Weight |
| 641 | • Height |
| 642 | |

# **Chapter 4: Follow-up Visits**

## 4.1 Follow-up Visits

- Follow-up Visits for all vision cohorts will occur annually. The Baseline Visit date is considered
- study day zero (0) from which follow-up visit windows are timed. The Follow-up Visit date will
- be the date the Follow-up Visit testing procedures started. All Follow-up Visit testing procedures
- will be completed on the same date other than the PROs as noted in **Section 4.4 Follow-up**
- 649 **Procedures**.

643

644

650

654

#### **4.2 Target Timelines**

- Target dates and windows for each study Follow-up Visit for all vision cohorts are shown below.
- Dates and windows are timed from Baseline Visit Date. Visits will be scheduled in the target
- window.

## Table 4-1. Schedule for Follow-up Visits

| VISIT SCHEDULE | TARGET DATE | TARGET WINDOW (AROUND TARGET DATE) |
|----------------|-------------|------------------------------------|
| 12 Month Visit | 52 Weeks | ± 4 Weeks |
| 24 Month Visit | 104 Weeks | ± 4 Weeks |
| 36 Month Visit | 156 Weeks | ± 4 Weeks |
| 48 Month Visit | 208 Weeks | ± 4 Weeks |

655 656

Table 4-2. Schedule for Remote Blood Spot Collection

| BLOOD SPOT<br>SCHEDULE | TARGET DATE | TARGET WINDOW (AROUND TARGET DATE) |
|------------------------|-------------|------------------------------------|
| 4 Months | 17 Weeks | ± 4 Weeks |
| 8 Months | 34 Weeks | ± 4 Weeks |
| 16 Months | 69 Weeks | ± 4 Weeks |
| 20 Months | 86 Weeks | ± 4 Weeks |
| 28 Months | 121 Weeks | ± 4 Weeks |
| 32 Months | 138 Weeks | ± 4 Weeks |
| 40 Months | 173 Weeks | ± 4 Weeks |
| 44 Months | 190 Weeks | ± 4 Weeks |

- The goal will be for all participants to complete all scheduled visits. However, participants who,
- because of unforeseen circumstances, are unable or unwilling to return for all follow-up visits
- will be permitted to return for key visits only as an alternative to withdrawal from the study.

| 660 | Additional office visits may occur as needed. |
|---|---|
| 661 | 4.3 Food Record and Blood Sample Collection |
| 662<br>663<br>664<br>665<br>666 | All participants will be asked to complete the blood sample collection as described below. Clinical Site Coordinators will complete a <b>Pre-Sample Collection Telephone Call</b> four (4) to ten (10) days prior to the scheduled sample collection date. For at-home samples, the <b>Post-Sample Collection Telephone Call</b> should be completed within one (1) day after the scheduled sample collection date. Reference the <b>GYROS Clinical Site Manual of Procedures</b> for more details. |
| 668 | (1) Participant Contact |
| 669 | <ul> <li>The Clinical Site Coordinator will contact the participants (via phone or other</li> </ul> |
| 670 | remote interface) four (4) to ten (10) days prior to the scheduled sample |
| 671 | collection date. The Pre-Sample Collection Telephone Call will include |
| 672 | instructions and reminders of: |
| 673 | <ul> <li>The next sample collection date.</li> </ul> |
| 674 | <ul> <li>Fasting instructions.</li> </ul> |
| 675 | o Food record collection instructions (if applicable; see Food Record |
| 676 | instructions below). |
| 677 | <ul> <li>For at-home sample collections the Clinical Site Coordinator will contact the</li> </ul> |
| 678 | participants (via phone or other remote interface) after the scheduled sample |
| 679<br>680 | collection date, within one (1) day preferred. The <b>Post-Sample Collection Telephone Call</b> will include the collection of: |
| 681 | o Information on the participant's last meal. |
| 682 | <ul> <li>Completion of the blood spot sample.</li> </ul> |
| 683 | <ul> <li>Completion of the Food Record.</li> </ul> |
| 684 | (2) Food Record |
| 685 | <ul> <li>Participants who indicated following an arginine-restricted diet at</li> </ul> |
| 686 | Screening will be asked to complete a food record every four (4) months |
| 687 | between Baseline and the 48M visit. |
| 688 | o If a participant initiates an arginine-restricted diet after Screening, the |
| 689 | participant will complete a food record every four (4) months going |
| 690 | forward. |
| 691 | <ul> <li>If a participant following an arginine-restricted diet at screening stops</li> </ul> |
| 692 | following an arginine-restricted diet at any point in the study, the |
| 693 | participant will continue to complete the food record every four (4) months. |
| 694<br>695 | <ul> <li>ALL participants will complete the food record for the 48M visit.</li> </ul> |
| 696 | The participants will complete the food record every day for three (3) days |
| 697 | prior to the fasting sample collection. |

| 698<br>699<br>700 | The participant will digitally send (e-mail or text) a picture of the food record to the site and either mail the original food record document to the site or bring it to the site at their next visit. |
|---|---|
| 701 | <ul> <li>The Clinical Site Coordinator will transcribe the data from the food record on the FFB Study Website.</li> </ul> |
| <ul><li>702</li><li>703</li><li>704</li><li>705</li></ul> | <ul> <li>A Central Dietitian Reviewer (CDR) will review food record on FFB Study Website to determine nutritional content. This information will be entered into the FFB Study Website.</li> </ul> |
| 706 | (3) Sample Collection |
| 707<br>708<br>709 | • At the annual Follow-up Visits, the Clinical Site Personnel will collect one (1) <u>fasting plasma sample</u> on all participants and ship to KKI. The sample collection procedures are detailed in the GYROS Clinical Site Manual of |
| 710 | Procedures. |
| 711<br>712<br>713 | • At the annual Follow-up Visits, the Clinical Site Personnel will collect one (1) <u>fasting blood spot fingerstick</u> on all participants and ship to KKI. The sample collection procedures are detailed in the GYROS Clinical Site Manual of Procedures. |
| 714<br>715<br>716<br>717 | <ul> <li>At the annual Follow-up Visits, the Clinical Site Coordinator would request the most recent lab records with an albumin result if the participant indicated they are <i>currently</i> on an arginine-restricted diet.</li> </ul> |
| 718<br>719<br>720<br>721<br>722<br>723 | ■ Every four (4) months between annual Follow-up Visits, one (1) <u>fasting</u> <u>blood spot fingerstick</u> will be collected on all participants. The participant or caretaker will collect the sample and ship to the central laboratory, KKI. The blood spot collection kits and instructions will be provided. The sample collection procedures are detailed in the GYROS Clinical Site Manual of Procedures. |
| 724 | 4.4 Follow-up Procedures |
| 725<br>726<br>727<br>728<br>729 | The following procedures will be performed at the Follow-Up Visits, unless otherwise specified. The testing procedures are detailed in the GYROS Clinical Site Manual of Procedures. An overview of the equipment and certification requirements for all testing is in <b>Chapter 5.1: Study Procedure Requirements</b> . All ocular testing will be performed in each eye, OD first and then OS. Follow-up visit procedures will last approximately seven (7) – eight (8) hours. |
| 730 | 4.4.1 Follow-up Data Collection and Testing Cohorts 1 & 2 |
| 731 | 1. Medical updates to include: |
| 732 | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 733 | <ul> <li>New ocular procedures</li> </ul> |
| 734 | <ul> <li>New or changed medications</li> </ul> |
| 735 | <ul> <li>Request medical records and laboratory records if applicable.</li> </ul> |
| 736 | 2. Patient Reported Outcomes |

| 737 | <ul> <li>Complete at 24-Month and 48-Month Follow-up Visits Only</li> </ul> |
|---|---|
| 738 | ◆ Adults: PROMIS®-29, MRDQ, ViSIO-PRO |
| 739 | <ul> <li>Adolescents: LPV-FVQ II, ViSIO-PRO</li> </ul> |
| 740 | <ul> <li>Children: LPV-FVQ II</li> </ul> |
| 741<br>742<br>743 | • The PROs may be completed in person or remotely (phone or other remote methods) any time within the Allowable Window of the associated visit, (not required to be the same day as the rest of the Follow up Visit). |
| 744 | 3. Complete ophthalmic examination to include: |
| 745 | Slit lamp biomicroscopy |
| 746 | <ul> <li>Indirect ophthalmoscopy</li> </ul> |
| 747 | <b>4.</b> IOP |
| 748 | • IOP measurements will be taken prior to pupil dilation. |
| 749 | 5. VA (including refraction, ETDRS, BRVT if needed, LLVA if needed) |
| 750<br>751<br>752 | <ul> <li>The visual acuity letter score will determine whether LLVA or BRVT will be<br/>performed. The criteria are defined in the GYROS Clinical Site Manual of<br/>Procedures.</li> </ul> |
| 753 | 6. SD-OCT |
| 754 | <ul> <li>Volume Scan</li> </ul> |
| 755 | <ul> <li>Vertical and Horizontal Scan</li> </ul> |
| 756 | 7. Axial Length and Corneal Curvature Measurements |
| 757 | <ul> <li>Complete at 24-Month and 48-Month Follow-up Visits Only</li> </ul> |
| 758 | 8. Fundus Autofluorescence |
| 759 | 9. Widefield color photo |
| 760 | <b>10.</b> OCTA |
| 761 | <ul> <li>Ancillary test; may be waived with approval from the Coordinating Center</li> </ul> |
| 762 | 11. Red reflex photo |
| 763 | 12. Full field Stimulus Threshold test (FST) |
| 764 | 13. Static perimetry |
| 765 | 14. Fundus guided microperimetry |
| 766 | 15. Measurements to include: |
| 767 | • Weight |
| 768 | • Height |
| 769 | <ul> <li>Measured annually in participants &lt;21 years of age at enrollment.</li> </ul> |

| 770 | 4.4.2 Follow-up Data Collection and Testing Cohort 3 |
|---|---|
| 771 | 1. Medical updates to include |
| 772 | <ul> <li>New or changed adverse events (AEs)</li> </ul> |
| 773 | <ul> <li>New ocular procedures</li> </ul> |
| 774 | <ul> <li>New or changed medications</li> </ul> |
| 775 | <ul> <li>Request medical records and laboratory records if applicable</li> </ul> |
| 776 | 2. Patient Reported Outcomes |
| 777 | <ul> <li>Complete at 24-Month and 48-Month Follow-up Visits Only</li> </ul> |
| 778 | ◆ Adults: PROMIS®-29, MRDQ, ViSIO-PRO |
| 779 | <ul> <li>Adolescents: LPV-FVQ II, ViSIO-PRO</li> </ul> |
| 780 | <ul> <li>Children: LPV-FVQ II</li> </ul> |
| 781<br>782<br>783 | <ul> <li>The PROs may be completed in person or remotely (phone or other remote<br/>methods) any time within the Allowable Window of the associated visit, (not<br/>required to be the same day as the rest of the Follow up Visit).</li> </ul> |
| 784 | 3. Complete ophthalmic examination to include: |
| 785 | <ul> <li>Slit lamp biomicroscopy</li> </ul> |
| 786 | <ul> <li>Indirect ophthalmoscopy</li> </ul> |
| 787 | <b>4.</b> IOP |
| 788 | <ul> <li>IOP measurements will be taken prior to pupil dilation.</li> </ul> |
| 789 | 5. VA (including refraction, ETDRS, BRVT if needed, LLVA if needed) |
| 790<br>791<br>792 | <ul> <li>The visual acuity letter score will determine whether LLVA or BRVT will be<br/>performed. The criteria are defined in the GYROS Clinical Site Manual of<br/>Procedures.</li> </ul> |
| 793 | 6. SD-OCT |
| 794 | <ul> <li>Volume Scan</li> </ul> |
| 795 | <ul> <li>Vertical and Horizontal Scan</li> </ul> |
| 796 | 7. Axial Length and Corneal Curvature Measurements |
| 797 | <ul> <li>Complete at 24-Month and 48-Month Follow-up Visits Only</li> </ul> |
| 798 | 8. Fundus Autofluorescence |
| 799 | 9. Widefield color photo |
| 800 | <b>10.</b> OCTA |
| 801 | <ul> <li>Ancillary test; may be waived with approval from the Coordinating Center</li> </ul> |
| 802 | 11. Red reflex photo |
| 803 | <b>12.</b> FST |

| 804 | 13. Measurements to include: |
|---|---|
| 805 | <ul><li>Weight</li></ul> |
| 806 | <ul> <li>Height</li> </ul> |
| 807 | <ul> <li>Measured annually in participants &lt;21 years of age at enrollment.</li> </ul> |
| 808 | 4.4.3 Unscheduled Visits |
| 809<br>810 | Testing procedures at unscheduled visits are at the investigator's discretion. However, it is recommended that procedures performed during these visits follow the standard protocol for |
| 811 | each procedure and be performed by certified personnel. Unscheduled visits will be recorded on |
| 812 | the FFB Consortium study website. Study images taken during unscheduled visits do not require |
| 813 | submission to the study website. |

# **Chapter 5: Testing Procedures and Questionnaires**

# **5.1 Study Procedure Requirements**

- The study procedure instructions are detailed in the **GYROS Clinical Site Manual of**
- Procedures. An overview of the equipment and certification requirements for all testing are
- provided in the table below.

815

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| Investigator taking overall responsibility for a visit | Oversees that consent process was performed in accordance with IRB/EC requirements; signs off on all eCRFs for a participant, eCRF edits, and protocol deviations. | N/A | Certified investigator |
| Coordinator taking responsibility for the visit | Oversees the data entry aspect of the visit; addresses protocol queries and signs off on deviations. | N/A | Certified coordinator |
| Informed Consent Form (ICF) Process | Explanation/review of study with the potential participant and/or signature of ICF. | N/A | Certified investigator as permitted by the IRB/EC |
| Signature of Informed<br>Consent Form | The participant and/or LAR sign the ICF. The person obtaining the ICF will also sign. | N/A | Certified investigator as permitted by the IRB/EC |
| Data entry on study website | Data collected from the study participant will be directly entered on the FFB Study Website (strongly encouraged) or written on the paper CRF and transcribed on the FFB Study Website within seven (7) days. | Computer and internet connection | Certified coordinator or certified investigator with additional study website certification |
| Collect information regarding medical history, demographics, adverse events, medications | Sites will collect medical history, demographic information, adverse events, and medications from the participant during each visit. This information can be confirmed by requesting medical records if needed. | N/A | Certified<br>investigator or<br>coordinator |
| Patient Reported<br>Outcomes | There will be a total of four (4) questionnaires. Three (3) for adults and one (1) – two (2) for minors depending on their age. | Study will provide | Certified investigator or coordinator |
| Ocular Exam | Including slit lamp biomicroscopy and indirect ophthalmoscopy | Any equipment is acceptable | Certified investigator |
| IOP | Measurement of the fluid pressure inside the eye. | Any equipment is acceptable | Clinical site personnel performing this test does not require a study |

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| | | | specific certification. However, they must be trained and delegated by the PI per the SSDL. |
| Visual Acuity – Refraction | Refraction is done as a routine part of<br>an eye exam to achieve best corrected<br>visual acuity measures | N/A | Clinical site<br>personnel<br>certified for<br>refraction |
| Visual Acuity – ETDRS | Traditional measure of central visual function that represents foveal cone function, | EVA system,<br>ETDRS charts | Clinical site<br>personnel<br>certified for<br>ETDRS |
| Visual Acuity – LLVA | LLVA tests vision function in low luminance conditions. | EVA system, or<br>ETDRS charts<br>2.0 neutral<br>density filter to<br>be provided by<br>study | Clinical site personnel certified for performing ETDRS is also certified to perform LLVA |
| Visual Acuity – BRVT | BRVT incorporates a three-level hierarchy for visual acuity testing better suited for low vision participants. | BRVT charts<br>provided by<br>study | Clinical site<br>personnel<br>certified for<br>BRVT |
| Spectral Domain Optical<br>Coherence Tomography -<br>Volume Scan | Scans provide objective, non-<br>invasive measures of retinal structure,<br>including loss of inner/outer segment<br>junction and have been shown to<br>correlate with visual function in eyes<br>with retinal degeneration | Heidelberg<br>Spectralis | Clinical site<br>personnel<br>certified for SD-<br>OCT |
| Spectral Domain Optical<br>Coherence Tomography -<br>Vertical and Horizontal<br>Scan | Scans provide objective, non-<br>invasive measures of retinal structure,<br>including loss of inner/outer segment<br>junction and have been shown to<br>correlate with visual function in eyes<br>with retinal degeneration | Heidelberg<br>Spectralis | Clinical site<br>personnel<br>certified for SD-<br>OCT and<br>vertical and<br>horizontal scan |
| ОСТА | Provides information on foveal<br>avascular zone enlargement and<br>decreased macular vascular density | Site must use pre-approved device. | Clinical site personnel certified for OCTA |
| Axial Length and Corneal<br>Curvature | Axial length measures the distance between the anterior and posterior poles of the eye. Corneal curvature determines the power of the cornea. | Any equipment is acceptable | Clinical site personnel performing this test does not require a study |

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| | | | specific certification. However, they must be trained and delegated by the PI per the SSDL. |
| Fundus Autofluorescence | Captures areas of absent<br>autofluorescence which corresponds<br>with areas of chorioretinal atrophy<br>seen on clinical exam | Optos | Clinical site<br>personnel<br>certified for<br>widefield fundus<br>autofluorescence |
| Widefield color photo<br>(UWF color) | Complementary imaging modality that delineates the borders of the atrophic lesions classically associated with GA | Optos | Clinical site<br>personnel<br>certified for<br>widefield color<br>photo |
| Red reflex photo | Captures the area and severity of posterior subcapsular cataracts commonly associated with GA | Digital camera capable of capturing external eye photos, Megapixels of >=3MP, Magnification of 30-40 degrees, Digital camera export in PNG, TIF, DICOM or BMP | Clinical site<br>personnel<br>certified for red<br>reflex photo |
| Full field Stimulus<br>Threshold test (FST) | Measures rod- and cone-mediated parts of the visual field | Diagnosys<br>Espion | Clinical site personnel performing this test does not require a study specific certification. However, they must be trained and delegated by the PI per the SSDL. |
| Static perimetry (SP) | A static field of vision test involves illuminating an object that does not move in the patient's field of vision to evaluate the vision in this manner. | Octopus 900<br>Pro (GATE<br>Protocol) | Clinical site<br>personnel<br>certified for SP |

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| Fundus guided<br>microperimetry (MP) | This test will map out how bright a spot needs to be for the participant to be see it at specific locations inside the eye. | MAIA | Clinical site<br>personnel<br>certified for MP |
| Kinetic Perimetry (KP) | A kinetic visual field test involves moving an object in and out of a patient's peripheral vision to find the edge of the patient's field of vision. | Any equipment is acceptable | Does not need to<br>be performed by<br>study certified<br>personnel or<br>recorded on the<br>GYROS Study<br>Staff Delegation<br>Log as this is a<br>historical test. |
| Three (3) day food record | A three-day food record is designed to get an accurate description of a participant's typical daily diet. | Source provided by the study | Certified investigator or coordinator |
| Blood sample collection: • Fasting plasma amino acids | The Amino Acids Analysis, Plasma is a blood test that measures 36 amino acids and intermediary metabolites. | N/A | Does not need to<br>be performed by<br>study certified<br>personnel or<br>recorded on the<br>GYROS Study<br>Staff Delegation<br>Log. |
| Blood sample processing: • Fasting plasma amino acids | During centrifugation, the barrier gel rises to separate the heavier cell mass from the lighter liquid portion. | Calibrated centrifuge | Certified investigator, coordinator, or appropriately trained laboratory staff |
| Measurements: Weight Height | Collect the participants height and weight using a calibrated scale in the office. BMI is automatically calculated on the FFB Study Website. | Calibrated scale | Certified investigator or coordinator |
| Skin Biopsy (3mm punch skin biopsy) | The skin is performed by stabilizing the area with the thumb and forefinger and stretched slightly perpendicular to the skin tension lines. A punch is held perpendicular to the skin, and is rotated into the skin with a firm, constant pressure. | Kit provided by the study | Certified investigator |
| Participant Contact<br>Reminders to complete the<br>three (3) day food record | The Clinical Site Coordinator will complete a <b>Pre-Sample Collection Telephone Call</b> to the participants (via phone or other remote interface) four (4) to ten (10) days prior to the scheduled sample collection date. | N/A | Certified investigator or coordinator |

| Study Procedures | Description | Equipment<br>Required<br>(If applicable) | Site Personnel<br>Delegation |
|---|---|---|---|
| | The Clinical Site Coordinator will complete a <b>Post-Sample Collection Telephone Call</b> for at-home samples within one (1) day after the scheduled sample collection date. | | |
| Food Record Collection<br>and transcription of data<br>on the FFB Study Website. | The Clinical Site Coordinator will collect and transcribe the data from the food record on the FFB Study Website | N/A | Certified investigator or coordinator |

# **5.2** Questionnaires

820

821 822 The following questionnaires will be administered in the study by a certified investigator or coordinator. Each questionnaire takes about fifteen (15) minutes to administer.

| Questionnaire | Туре | Description | Vision<br>Cohort | Age |
|---|---|---|---|---|
| Michigan Retinal<br>Degeneration<br>Questionnaire<br>(MRDQ) | Vision<br>Function | The MRDQ is a psychometrically validated patient-reported outcome measure for inherited retinal degenerations questionnaire which consists of fifty-nine (59) questions measuring seven (7) unidimensional domains: central vision, color vision, contrast sensitivity, scotopic function, photopic peripheral vision, and photosensitivity. | All | Adults >= 18<br>years |
| PROMIS-29®<br>(Patient-Reported<br>Outcomes<br>Measurement<br>Information<br>System®) | Global physical, mental, and social health | The PROMIS®-29 contains items from seven PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. The seven domains cover the most relevant areas of self-reported health for most people with chronic illness. There is also one 11-point rating scale for pain intensity. | All | Adults >= 18<br>years |
| Visual Symptom<br>and Impact<br>Outcomes Patient<br>Reported Outcome<br>(ViSIO-PRO) | Vision<br>Function<br>and<br>HRQoL | The ViSIO-PRO is an instrument designed to assess visual function symptoms, impacts on functional vision, and impacts on wider health-related quality of life (HRQoL). It has been designed for completion by adolescents (12-17) and adults (18 +) with retinitis pigmentosa (RP). | All | Adolescents<br>(12-17) and<br>Adults (18+) |
| L. V. Prasad-<br>Functional Vision | Vision<br>Function | The LVP-FVQ-II questionnaire consists of twenty-three (23) | All | Children<br>(<18 years) |

| Questionnaire<br>(LVP-FVQ II) | questions. The questionnaire is used to assess self-reported difficulties in |
|---|---|
| | performing daily tasks in children with visual impairment. |

#### **Chapter 6: Unanticipated Problem and** 824 **Adverse Event Reporting** 825 **6.1 Unanticipated Problems** 826 Site investigators will promptly report all unanticipated problems meeting the criteria below on 827 an eCRF. Sites overseen by the JCHR IRB must report Unanticipated Problems to the IRB 828 within seven (7) calendar days of recognition. For this protocol, an unanticipated problem is an 829 incident, experience, or outcome that meets all the following criteria: 830 • Unexpected (in terms of nature, severity, or frequency) given (a) the research 831 procedures that are described in the protocol related documents, such as the IRB-832 approved research protocol and informed consent document; and (b) the 833 characteristics of the subject population being studied. 834 • Related or possibly related to participation in the research (possibly related means 835 there is a reasonable possibility that the incident, experience, or outcome may have 836 been caused by the procedures involved in the research). 837 • Suggests that the research places participants or others at a greater risk of harm than 838 was previously known or recognized (including physical, psychological, economic, or 839 social harm). 840 The CC will report to the IRB all unanticipated problems not directly involving a specific site 841 842 such as unanticipated problems that occur at the CC or at another participating entity such as a laboratory. 843 These instances must be reported to the JCHR IRB within seven (7) calendar days of recognition. 844 The Director of the Human Research Protection Program (HRPP) will report to the appropriate 845 regulatory authorities and applicable relying IRBs if the JCHR IRB determines that the event 846 indeed meets the criteria of an Unanticipated Problem that requires further reporting to fulfill the 847 reporting obligations of the HRPP. 848 **6.2 Adverse Events** 849 6.2.1 Definitions 850 Adverse Event (AE): Any untoward medical occurrence, including laboratory findings, 851 associated with study procedures whether the event is considered related. Progression of GA 852 retinal dystrophy including new or worsening of anticipated clinical signs or symptoms, which 853 are collected and assessed as unequivocally associated with the disease progression should NOT 854 be reported as AEs unless the disease progression is greater than anticipated in the natural course 855 of the disease. 856 Serious Adverse Event (SAE): Any untoward medical occurrence that results in any of the 857 following outcomes: 858 • Death. 859 • A life-threatening adverse event: (a non-life-threatening event which, had it been 860 more severe, might have become life-threatening, is not necessarily considered a 861 serious adverse event). 862

- \* Inpatient hospitalization or prolongation of existing hospitalization.
  - A persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions.
    - A congenital anomaly or birth defect.
- An important medical event that may not result in death, be life-threatening, or require
- hospitalization may be considered serious when, based upon appropriate medical judgment, they
- may jeopardize the patient or subject and may require medical and surgical intervention to
- prevent one of the outcomes listed in this definition.
- Note: As this is a Natural History Study, the Investigator(s) will make the categorical
- determinations of Adverse Events, as described above, and will report each determination to the
- 873 Coordinating Center, as per data collection.

#### **6.2.2 Reportable Adverse Events**

- For this protocol, a reportable adverse event includes all events meeting the definition of an
- adverse event.

864

865

866

874

885

- All reportable Adverse Events whether volunteered by the participant, discovered by study
- personnel during questioning, or detected through ophthalmological examination, laboratory test,
- or other means will be reported on an adverse event form online.
- The purpose of AE collection for the GYROS study will be to provide historical controls for
- future clinical trials. As a no greater than minimal risk study, AEs do not require any specific
- reporting to regulatory or oversight bodies. However, each Principal Investigator is responsible
- for abiding by any other reporting requirements specific to their IRB or equivalent ethics
- 884 oversight committee

#### 6.2.3 Relationship of Adverse Event to Study Procedure

- The study investigator will assess the relationship of any adverse event to be related or unrelated
- to a study procedure by determining if there is a reasonable possibility that the adverse event
- may have been caused by the study procedure.
- To ensure consistency of adverse event causality assessments, investigators should apply the
- following general guideline when determining whether an adverse event is related:
- 891 **Yes**
- There is a plausible temporal relationship between the onset of the adverse event and the study
- procedure, and the adverse event cannot be readily explained by the participant's clinical state,
- intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern
- of response to the study procedure; and/or the adverse event abates or resolves upon
- 896 discontinuation of the study procedure.
- 897 **No**
- 898 Evidence exists that the adverse event has an etiology other than the study procedure (e.g.,
- 899 preexisting medical condition, underlying disease, intercurrent illness, or concomitant
- medication); and/or the adverse event has no plausible temporal relationship to study procedure.

#### 6.2.4 Severity (Intensity) of Adverse Event 901 A severity assessment is a clinical determination of the intensity of an event. Thus, a severe 902 adverse event is not necessarily serious. For example, itching for several days may be rated as 903 severe, but may not be clinically serious. 904 The severity (intensity) of an adverse event will be rated on a three-point scale: (1) mild, (2) 905 moderate, or (3) severe. 906 907 1. MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily activities. 908 909 2. MODERATE: Usually causes a low level of inconvenience, discomfort or concern to the participant and may interfere with daily activities but is usually ameliorated by 910 simple therapeutic measures and participant is able to continue in study. 911 3. SEVERE: Interrupts a participant's usual daily activities and causes severe 912 discomfort. 913 6.2.5 Expectedness 914 As this is a Natural History Study, the expectedness for a serious adverse event will not be 915 916 assessed. **6.2.6 Coding of Adverse Events** 917 Adverse events will be coded using the MedDRA dictionary. To facilitate coding, the site will 918 enter a preliminary MedDRA code 919 6.2.7 Outcome of Adverse Event 920 The outcome of each reportable adverse event will be classified by the investigator as follows: 921 1. RECOVERED/RESOLVED (COMPLETE RECOVERY) – The participant 922 recovered from the AE/SAE without sequelae. Record the AE/SAE stop date. 923 2. RECOVERED/RESOLVED WITH SEQUELAE – AE/SAE where the subject 924 recuperated but retained pathological conditions resulting from the prior disease or 925 injury. Record the AE/SAE stop date. 926 3. FATAL – A fatal outcome is defined as the SAE that resulted in death. Only the 927 event that was the cause of death should be reported as fatal. AEs/SAEs that were 928 ongoing at the time of death; however, were not the cause of death, will be recorded 929 as "resolved" at the time of death. 930 4. ONGOING NOT RECOVERED/NOT RESOLVED – An ongoing AE/SAE is 931 defined as an ongoing event with an undetermined outcome. 932 An ongoing outcome will require follow-up by the site to determine the outcome 933 of the AE/SAE. 934 The outcome of an ongoing event at the time of death that was not the cause of 935 death, will be updated and recorded as "resolved" with the date of death recorded 936

937

as the stop date.

| 938<br>939 | <b>5. ONGOING (MEDICALLY STABLE)</b> – AE/SAE is ongoing, but medically stable. For example, a chronic condition where no further change is expected. |
|---|---|
| 940<br>941<br>942<br>943<br>944 | If any reported adverse events are ongoing when a participant completes the study (or withdraws), they will be followed until they are either resolved, or have no prospect of improvement or change, even after the participant has completed all applicable study visits/contacts. For all other adverse events, data collection will end at the time the participant completes the study. |
| 945<br>946 | <b>Note:</b> participants should continue to receive appropriate medical care for an adverse event after their participation in the study ends. |
| 947<br>948 | If a participant is lost to follow up and participant outcome cannot be determined, outcome classification will be the last known outcome. |
| 949 | 6.3 Timing of Event Reporting |
| 950<br>951 | Investigator(s) are responsible for reporting Adverse Events on the electronic case report form (eCRF) through the study website in a timely manner. |
| 952<br>953<br>954<br>955<br>956 | Each Principal Investigator (PI) is responsible for reporting serious study-related adverse events and abiding by any other reporting requirements specific to his/her Institutional Review Board (IRB) or Ethics Committee (EC). Where the JCHR IRB is the overseeing IRB, sites must report all serious, related adverse events regardless of whether they are expected/anticipated and regardless of whether they are fatal or life-threatening within seven (7) calendar days. |
| 957 | |

#### **Chapter 7: Miscellaneous Considerations** 958 7.1 New or ongoing Medical Conditions and Medications 959 7.1.1 Pre-Existing Condition 960 Any medical condition that is either present at screening, a chronic disease, or a prior condition 961 that could impact the participant's health during the study (e.g., prior myocardial infarction or 962 stroke). 963 7.1.2 Medical Conditions during the study 964 In addition to conditions meeting the reporting requirements for an adverse event or as described 965 above, the following medical conditions should also be reported: (1) new diagnosis of a chronic 966 disease (i.e., not present at the time of enrollment), and (2) any medical condition that could 967 affect the participant's ability to carry out any aspect of the protocol or could affect an outcome 968 assessment. These will be reported as adverse events. See Chapter 6.2 Adverse Events for more 969 detail. 970 7.1.3 Medications 971 All medication for the treatment of chronic pre-existing conditions, medical conditions, and/or 972 adverse events that the participant is currently taking at screening and during the study should be 973 recorded. Nutraceuticals and preventative treatments that are of interest to the study will be 974 975 recorded. 7.2 Prohibited Medications, Treatments, and Procedures 976 7.2.1 Prohibited Medications and Treatment for *OAT*-Related Retinal Degeneration 977 Participants who are **enrolled into the final study cohort** should not receive IRD treatments 978 during the study. This includes enrolling into an experimental treatment trial of underlying 979 980 conditions related to OAT mutations during the 4-year study duration. However, if the participants enroll in a treatment trial the Executive Committee will be consulted and will 981 determine if the participant may continue in the study. 982 Examples of prohibited medications and treatments include, but are not limited to the following: 983 • use of ocular stem cell or gene therapy 984 ocriplasmin 985 ophthalmic oligonucleotide 986 Ozurdex (dexamethasone) 987 • Iluvien or 988 Yutiq (fluocinolone acetonide) intravitreal implant 989 Amiodarone, chloroquine, deferoxamine, hydroxychloroquine, pentosan polysulfate, 990 tamoxifen, thioridazine 991

#### 7.2.2 Intraocular Surgical Procedures 992 Participants enrolled into the final study cohort, who have intraocular surgery during the study, 993 will have follow-up visits timed either before the surgery date or at least three (3) months after 994 the surgery date. Clinical sites will make reasonable efforts to schedule the participant's follow-995 up visit as close to the visit target window as possible. 996 7.2.3 Treatment for Cystoid Macular Edema (CME) 997 Participants enrolled into the final study cohort, who need to receive treatment for CME 998 during the study, may do so with an oral or topical dorzolamide, topical nonsteroidal or 999 injectable corticosteroid, but not a steroid implant. 1000 7.3 Pregnancy Reporting 1001 If a pregnancy occurs, the participant will remain in the study. The occurrence of pregnancy will 1002 be reported to the Coordinating Center within seven (7) days of the site's discovery of the 1003 pregnancy (including at screening) and the Pregnancy Notification form will be completed 1004 within seven (7) calendar days. Sites will collect concomitant medications throughout the 1005 pregnancy. If an Adverse Event occurs because of the pregnancy, then the site will record the 1006 Adverse Event on the Adverse Event form. 1007 7.4 Participant Compensation 1008 Participant compensation will be specified in the informed consent form. 1009 7.5 Participant Withdrawal 1010 Participation in the study is voluntary, and a participant may withdraw at any time. For 1011 participants who withdraw, their data will be used up until the time of withdrawal. 1012 7.6 Confidentiality 1013 For security and confidentiality purposes, participants will be assigned an identifier that will be 1014 used instead of their name. Protected health information gathered for this study will be shared 1015

with the coordinating center, the Jaeb Center for Health Research in Tampa, FL. De-identified

participant information may also be provided to research sites involved in the study.

1016

# **Chapter 8: Statistical Considerations**

## 8.1 Statistical and Analytical

The approach to sample size and statistical analyses are summarized below. The analysis plan synopsis in this chapter contains the framework of the anticipated final analysis plan.

#### 8.2 Sample Size

 The sample size evaluation focuses on objective 1a of the study, to characterize the natural history of retinal degeneration associated with disease-causing *OAT* variants in the presence of standard care dietary treatment regimens over four (4) years, using functional, structural, and patient-reported outcome measures. A justification of the selected sample size using percent change for the outcomes of interest is outlined. The precision of estimates and of the correlation between structure-based, function-based, and metabolic-based outcomes involved in objective two (2) and of the correlation between eyes in the outcomes is also provided. Calculations to address objective three (3), explore risk factors associated with progression (i.e., compare subgroups for dichotomous risk factors), are summarized.

# 8.2.1 Sample Size Considerations for Evaluating Percent Change from Baseline to four(4) Years – All Outcomes

Longitudinal changes on all outcome parameters being collected will be examined with the change in preserved retina being of particular interest. Change from baseline to four (4) years will be evaluated for sample size purposes, although statistical analyses will include the data from each annual visit. The power and sample size calculations below may be used to consider percent change on any outcome measure from baseline to four (4) years.

Both eyes of a participant will be assessed for the main outcomes of interest. Thus, if there are N participants, 2N eyes will be available for analysis. However, outcome measures from two (2) eyes of a person are typically strongly correlated ( $r \ge 0.5$ ). The contribution of information from the two (2) eyes in this case is (2/(1+r)) instead of two (2). Values for the multiplier to the number of participants to obtain an effective sample size are given below:

| Effective<br>N |
|----------------|
| 2.00 |
| 1.82 |
| 1.67 |
| 1.54 |
| 1.43 |
| 1.33 |
| 1.25 |
| 1.18 |
| 1.11 |

| 0.9 | 1.05 |
|-----|------|
| 1.0 | 1.00 |

The correlation between eyes (inter-eye correlation) for each outcome measure will be estimated during the study and is not known at the time of study design. We assume here a correlation of 0.8. This assumption is conservative in that it requires a higher number of participants than lower plausible values of r.

The primary way sample size is evaluated is by considering the precision around the point estimates for the percent change in the outcome measures over four (4) years. **Table 6.1** provides the half width of the 95% confidence interval (CI) for the estimated mean percent change per year for combinations of the standard deviation (SD) of the distribution of percent change and sample size. The larger the SD, the wider the CI, meaning the range of possible true values grows.

Table 6.1. Sample size versus half width of 95% confidence interval for the mean percent change for varying standard deviation values.

| | Effective Sample Size (N of participants) | | | | |
|---|---|---|---|---|---|
| | n=11 (10) | n=11 (10) | | | |
| SD=20% | 12% | 8% | 7% | 6% | 5% |
| SD=30% | 18% | 13% | 10% | 9% | 8% |
| SD=40% | 24% | 17% | 14% | 12% | 11% |
| SD=50% | 30% | 21% | 17% | 15% | 13% |

Note: The shaded column corresponds to the sample size deemed feasible based on preliminary patient counts and financial constraints. Forty (40) participants from Vision Cohorts 1 and 2 will be followed for progression.

# 8.2.2 Sample Size Considerations for Comparing Percent Change from Baseline to four (4) Years within Subgroups of Interest – All Outcomes

Another objective for this natural history study will be to explore the association of risk factors with progression of various functional outcome variables (objective 3). **Figure 6.1** considers various expected SDs of the distribution of percent change from baseline to four (4) years per eye and evaluates the power to detect varying differences in average percent change from baseline to four (4) years, comparing subgroups of various equally distributed sizes. If subgroups are not equally sized the smallest detectable difference (with the same power) will be larger. Testing will be performed with a Type I ( $\alpha$ ) error rate of 0.05.

**Note:** <u>within</u> subgroup point estimates and Cis will also be important. **Table 6.1** above can be applied to potential subgroup sample sizes as well to consider the precision that would be observed.



Figure 6.1. Power to conclude there is a difference given varying true difference values, population standard deviation, and sample size.

For the graphs is Figure 6.1, the y-axis if for the power to conclude that there is a difference when the true difference in mean percent change is the x-axis value. Each of the four graphs is for a different total sample size with the number of eyes in each of the two subgroups being approximately fifty percent (50%). Forty (40) participants from Vision Cohorts 1 and 2 will be followed.

For example, with an effective sample size of twenty-two (22) and an effective sample size of eleven (11) in each subgroup, to have power of 80% or more, the true difference needs to be approximately 1.25 SDs (a mean difference of 25% if the SD of the percent change over four (4) years 20%). If the effective sample size is thirty-three (33), the true difference needs to be approximately 1.0 SD (a mean difference 20% if the SD of the percent change over four (4) years is 20%). If the effective sample size is forty-four (44), the true difference needs to be approximately 0.86 SDs (a mean difference 17% if the SD of the percent change over four (4) years is 20%). Such mean differences are considered large.

# 8.2.3 Sample Size Considerations for Precision of the Estimate of the Correlation Between Structure-based, Function-based, and Metabolic-based Outcomes and of the Correlation Between Eyes

The Pearson correlation coefficient (r) can be used to assess the correlation between two different outcome measures. The distribution of r is not symmetric; therefore, CIs for the estimated correlation coefficient are not symmetric. A transformation of r (z = 0.5 \* ln ((1+r)/1-r)) is used to create a variable that is asymptotically distributed N (0, 1/(sqrt(N-3))) under the null hypothesis that r=0.

The intraclass correlation coefficient is used to assess the strength of agreement between eyes. When both eyes have the same mean for the outcome measure, the intraclass correlation coefficient is equal to the standard Pearson correlation coefficient (r). The table below provides the 95% CI for different estimates of r from the observed data.

Table 6.2A. 95% Confidence Intervals for an Observed Value of the Correlation between Outcome Measures.

| | Effective sample size | | | | |
|---|---|---|---|---|---|
| r | n= 11 | n= 22 | n= 33 | n= 44 | n=55 |
| 0.3 | (-0.37,0.76) | (-0.14,0.64) | (-0.05,0.58) | (0.00,0.55) | (0.04,0.52) |
| 0.4 | (-0.26,0.81) | (-0.03,0.70) | (0.07,0.65) | (0.12,0.62) | (0.15,0.60) |
| 0.5 | (-0.14,0.85) | (0.10,0.76) | (0.19,0.72) | (0.24,0.69) | (0.27,0.68) |
| 0.6 | (0.00,0.88) | (0.24,0.82) | (0.32,0.78) | (0.37,0.76) | (0.40,0.75) |
| 0.7 | (0.17,0.92) | (0.39,0.87) | (0.47,0.84) | (0.51,0.83) | (0.53,0.81) |
| 0.8 | (0.38,0.95) | (0.57,0.91) | (0.63,0.90) | (0.66,0.89) | (0.68,0.88) |
| 0.9 | (0.65,0.97) | (0.77,0.96) | (0.81,0.95) | (0.82,0.94) | (0.83,0.94) |

Table 6.2B. 95% Confidence Intervals for an Observed Value of the Inter-eye Correlation.

| | N of patients | | | | |
|---|---|---|---|---|---|
| r | n= 10 | n= 20 | n= 30 | n= 40 | n=50 |
| 0.3 | (-0.41,0.78) | (-0.16,0.66) | (-0.07,0.60) | (-0.01,0.56) | (0.02,0.53) |
| 0.4 | (-0.31,0.82) | (-0.05,0.72) | (0.05,0.66) | (0.10,0.63) | (0.14,0.61) |
| 0.5 | (-0.19,0.86) | (0.07,0.77) | (0.17,0.73) | (0.22,0.70) | (0.26,0.68) |
| 0.6 | (-0.05,0.89) | (0.21,0.82) | (0.31,0.79) | (0.35,0.77) | (0.39,0.75) |
| 0.7 | (0.13,0.92) | (0.37,0.87) | (0.45,0.85) | (0.50,0.83) | (0.52,0.82) |
| 0.8 | (0.34,0.95) | (0.55,0.92) | (0.62,0.90) | (0.65,0.89) | (0.67,0.88) |
| 0.9 | (0.62,0.98) | (0.76,0.96) | (0.80,0.95) | (0.82,0.95) | (0.83,0.94) |

1086

1087

1088

1094

1095

1096

10971098

1099

Note: The shaded column corresponds to the sample size deemed feasible based on preliminary patient counts

and financial constraints. Forty (40) participants from Vision Cohorts 1 and 2 will be followed and used for

Longitudinal changes in all outcome parameters being collected will be of interest for objectives

one (1) and three (3). Information on rates of decline using the proposed outcome measures for

• Valproic Acid Protocol (VPA) Data (phase II multiple sites, randomized, placebo-

controlled trial of oral valproic acid for ADRP) [Placebo group N=44; dataset can be

• Expect average annual decline due to *OAT* will be 5% per year or 20% by four (4) years.

• True SD of percent change at four (4) years is like VPA 1-year SD of approximately

OAT variants does not exist. 12,26 Information on rates of decline for inherited retinal

o Percent Change from Baseline to 1 year, Mean (SD):

assessing inter-eye correlation of change in outcome measures over time.

**8.2.4** Final Sample Size Justification

Data to consider for evaluating sample size:

accessed at https://public.jaeb.org/ffb/stdy]

-0.3% (16%) OD

-4.9% (17%) OS

degenerations in general is limited.

**Assumptions made:** 

20%. 1119 1120 If thirty (30) study participants or thirty-three (33) effective eyes are recruited: 1121 • The half width of a 95% CI around the point estimate for mean percent change would be 1122 1123 seven (7) %. A comparison of two equal-sized subgroups would have about 80% power to conclude 1124 1125 there is a difference if the true difference is 20%. For the objective of evaluating the agreement in outcome between eyes, a sample size of 1126 thirty (30) participants for Vision Cohorts 1 and 2 will yield a 95% CI of (0.17,0.73) 1127 when the observed r equals 0.5, and (0.62,0.90) when the observed r equals 0.8. 1128 • For the objective of evaluating the correlation between outcomes, an effective sample 1129 size of thirty-three (33) participants for Vision Cohorts 1 and 2 will have a 95% CI of 1130 (0.19,0.72) when the observed r equals 0.5, and (0.63,0.90) when the observed r equals 1131 0.8. 1132 1133 If forty (40) study participants or forty-four (44) effective eyes are recruited: 1134 • The half width of a 95% CI around the point estimate for mean percent change would be 1135 six (6) %. 1136 • A comparison of two equal-sized subgroups would have about 80% power to conclude 1137 there is a difference if the true difference is 17%. 1138 • For the objective of evaluating the agreement in outcome between eyes, a sample size of 1139 forty (40) participants for Vision Cohorts 1 and 2 will yield a 95% CI of (0.22,0.70) when 1140 the observed r equals 0.5, and (0.65,0.89) when the observed r equals 0.8. 1141

1101 1102

1103

1104

1105

1106

1107

1108

1109

1110 1111

1112

1113

1114 1115

1116

1117

• For the objective of evaluating the correlation between outcomes, an effective sample size of forty-four (44) participants for Vision Cohorts 1 and 2 will yield a 95% CI of (0.24,0.69) when the observed r equals 0.5, and (0.66,0.89) when the observed r equals 0.8.

#### 8.3 Data Analysis

The analysis plans below are written with respect to most outcomes of interest. Analyses will include data on both eyes for each participant, and confidence intervals will be adjusted for correlation between two (2) eyes of the same participant.

#### 8.3.1 Primary Objective Analysis

The primary objectives of the natural history study and brief analysis plan for each are as follows.

#### 1. Natural History

- (a) Characterize the natural history of retinal degeneration associated with disease-causing *OAT* variants over four (4) years, as measured using functional, structural, and patient-reported outcome measures.
  - i. Functional and structural measures: The distribution of each outcome at each visit will be summarized (including tabulating categorically, as well as means, SDs, medians, quartiles, ranges; both the absolute change and percent change will be evaluated, tests performed multiple times per visit will be analyzed using the average of all available tests). To determine the average annual rate of progression in the population for each outcome, a mixed effects model will be fit using all available outcome data at baseline and all annual visits. Both the correlation in outcomes over time and the correlation in outcomes between eyes will be accommodated by the model.<sup>28</sup> Mixed models adequately accommodate missing values when missing values are missing at random (MAR). A second method of accommodating missing values will be through multiple imputation for the outcome values for all missing time points (including participants who discontinue follow up prior to forty-eight (48) months). Secondary analyses using binary definitions of outcome measures will also be explored in time to event analyses; Kaplan-Meier estimates with 95% confidence intervals will be calculated.
  - ii. PRO measures: The scoring of each questionnaire will be completed according to the procedures recommended by the developers of the questionnaire for each instrument. Baseline scores will be cross tabulated with categorical (severity of disease) versions of the outcome measures of interest at baseline. Changes in scores will be cross tabulated with binary (progression of disease) versions of the outcome measures of interest at the 24- and 48-month visits. A generalized linear model adjusted for baseline differences will be explored.

1146

1150

1151

1152

1153

1154

117511761177

1178

1179

1180

1181

1182

1183

| 1185 | Partially completed questionnaires will be managed using methods |
|---|---|
| 1186 | recommended by the developers of the specific questionnaire. When |
| 1187 | no questionnaire is completed, we will use statistical methods that |
| 1188 | mitigate the impact of missing data, specifically, mixed effects |
| 1189 | regression models and multiple imputation for the outcome values for |
| 1190 | all missing time points. |
| 1191 | |
| 1192 | (b) Characterize the natural history of ornithine levels associated with disease- |
| 1193 | causing <i>OAT</i> variants in the presence of standard care dietary treatment |
| 1194 | regimens over four (4) years. |
| 1195 | |
| 1196 | i. Longitudinal annual measures of ornithine will be explored by |
| 1197 | graphing the values for everyone ("spaghetti" plots) and analyzed to |
| 1198 | detect any linear trend in time with mixed effects models. |
| 1199 | · |
| 1200 | (c) Determine within-patient variability of ornithine levels associated with |
| 1201 | disease-causing <i>OAT</i> variants in the presence of standard care dietary |
| 1202 | treatment regimens over four (4) years. |
| 1203 | i. The within-person standard deviation of ornithine levels will be |
| 1204 | estimated for the group of patients using a mixed effects model. |
| 1205 | Models will be based on levels from blood dot tests and from plasma |
| 1206 | testing over the four (4) years to determined long -term variability and |
| 1207 | on levels from blood dot tests over periods of six (6) months and of |
| 1208 | twelve (12) months to determine short-term variability. The coefficient |
| 1209 | of repeatability will be calculated to estimate the difference from |
| 1210 | baseline that would need to be exceeded to indicate that a treatment |
| 1211 | was causing an effect beyond random variability. |
| 1212 | 2. Metabolic, Structure, and Function Relationships |
| 1213 | (a) Evaluate cross-sectional associations at baseline and each annual visit with |
| 1214 | scatterplots and Spearman correlation coefficients. Evaluate the association of |
| 1215 | changes in each outcome measure with changes the other outcome measures |
| 1216 | at each visit with scatter plots and Spearman correlation coefficients. Use |
| 1217 | mixed effects regression models to evaluate the association of change in each |
| 1218 | outcome measure with changes in each of the other outcome measures. With |
| 1219 | so many outcomes and only forty (40) patients, results will be interpreted |
| 1220 | cautiously because of both low powers to detect clinically meaningful |
| 1221 | associations and elevated Type I error rates due to multiple comparisons. |
| 1222 | 3. Identify Rapid Progressors |
| 1223 | (a) The distribution of each outcome in terms of both absolute change and percent |
| 1224 | change from baseline to four (4) years will be summarized (including |
| 1225 | tabulating categorically, as well as means, standard deviations, medians, |
| 1226 | quartiles), stratified by categorical levels of each potential risk factor of |
| 1227 | interest (listed below). Potential risk factors to evaluate include phenotypic |
| 1228 | factors including the baseline level of each of the structural and functional |

| 1229 | measures and ornithine level, genotype, and adherence to the arginine- |
|---|---|
| 1230 | restricted diet as noted below. Univariable regression models of each outcome |
| 1231 | measure will be fit for each of the potential risk factors. With so many |
| 1232 | potential risk factors and outcomes and only forty (40) patients, results will be |
| 1233 | interpreted cautiously because of both low powers to detect clinically |
| 1234 | meaningful differences and elevated Type I error rates due to multiple |
| 1235 | comparisons. |
| 1236 | |
| 1237 | i. Phenotypic: |
| 1238 | <ul> <li>Age of onset of initial vision symptoms</li> </ul> |
| 1239 | <ul><li>Gender</li></ul> |
| 1240 | <ul><li>Race/ethnicity</li></ul> |
| 1241 | <ul> <li>Body weight/BMI</li> </ul> |
| 1242 | <ul> <li>Lens Status (phakic/pseudophakic/aphakic) and area of</li> </ul> |
| 1243 | subcapsular cataract on red reflex photos |
| 1244 | <ul> <li>Baseline foveal avascular zone (FAZ) area and macular vessel</li> </ul> |
| 1245 | density on OCTA |
| 1246 | <ul> <li>Baseline visual acuity</li> </ul> |
| 1247 | <ul> <li>Baseline low luminance visual acuity</li> </ul> |
| 1248 | <ul> <li>Baseline area of preserved retina on fundus autofluorescence</li> </ul> |
| 1249 | and color photos |
| 1250 | <ul> <li>Baseline full Hill of Vision (HOV) on static perimetry</li> </ul> |
| 1251 | <ul> <li>Baseline mean sensitivity on static perimetry</li> </ul> |
| 1252 | <ul> <li>Baseline mean retinal sensitivity on microperimetry</li> </ul> |
| 1253 | <ul> <li>Baseline full-field stimulus (FST) levels</li> </ul> |
| 1254 | <ul> <li>Baseline ERG amplitude and timing</li> </ul> |
| 1255 | <ul> <li>Baseline ellipsoid zone (EZ) area on OCT</li> </ul> |
| 1256 | <ul> <li>Baseline ornithine level</li> </ul> |
| 1257 | |
| 1258 | ii. Genotypic |
| 1259 | • Characterizations of the <i>OAT</i> variants |
| 1260 | |
| 1261 | iii. Environmental Factors |
| 1262 | <ul> <li>Adherence to arginine-restricted diet</li> </ul> |
| 1263 | <ul><li>Smoking</li></ul> |
| 1264 | C C C C C C C C C C C C C C C C C C C |

#### **Chapter 9: Data Collection and Monitoring** 1265 9.1 Case Report Forms and Other Data Collection 1266 The main study data are collected on electronic case report forms (eCRFs). When data are 1267 directly collected in electronic case report forms, this will be considered the source data. 1268 However, it is recommended that a progress note is completed to document the events of the 1269 visit. For any data points for which the eCRF is not considered source (e.g., lab results that are 1270 transcribed from a printed report into the eCRF), the original source documentation must be 1271 maintained in the participant's study chart or medical record. This source must be readily 1272 verifiable against the values entered into eCRF. Even where all study data are directly entered 1273 into the eCRFs at office visits, evidence of interaction with a live subject must be recorded (e.g., 1274 office note, visit record, etc.) and provided to the coordinating center for review. 1275 Each participating site will maintain appropriate medical and research records for this trial, in 1276 compliance with International Council for Harmonisation of Technical Requirements for 1277 Pharmaceuticals for Human Use (ICH) E6 and regulatory and institutional requirements for the 1278 protection of confidentiality of participants. 1279 9.1.1 Central Lab 1280 The Kennedy Krieger Institute, Central Lab, will complete an analysis from the fasting amino 1281 acid panel, and blood spot collection. The lab will directly enter the laboratory results on the FFB 1282 Study Website. 1283 Results for ornithine and arginine will be provided for the site. 1284 1285 9.1.2 Research Lab The Johns Hopkins University Department of Genetic Medicine Research Lab will receive the 1286 skin biopsy samples to grow fibroblasts. The tissue sample analysis will be entered directly in the 1287 FFB Study Website. 1288 9.1.3 Central Genetics Auditor (CGA) 1289 The CGA will review the genetic lab report(s) submitted by the clinical site during genetic 1290 screening against the genetic eCRF data to ensure that the data entered by the clinical site are 1291 consistent with the source(s) provided prior to the Baseline visit. The CGA will document his/her 1292 verification of these genetic data on the FFB Consortium study website and the clinical site will 1293 be notified of the results of the review. 1294 9.1.4 Genetics Committee 1295 In addition to providing evaluation of whether the *OAT* mutations are causative of the disease on 1296 the FFB Consortium study website, the Genetics Committee will review and provide approval 1297 for the use of genetic reports from research labs to be used for determining participant eligibility. 1298

| 1299<br>1300 | 9.1.5 The Johns Hopkins Institute for Clinical and Translational Research (ICTR) Research Nutrition |
|---|---|
| 1301<br>1302<br>1303<br>1304 | The site will enter the food record documentation on the FFB Study Website. ICTR will review the three (3) day food records and analyze for arginine, vitamin A, and vitamin B6 intake. Total protein and caloric intake will be documented as well. ICTR will enter the nutrition analysis assessment data directly on the FFB Study Website. |
| 1305 | 9.1.6 Reading Centers |
| 1306<br>1307<br>1308<br>1309 | Reading Centers will conduct grading of the study data collected using the FFB Consortium study website. The Reading Centers will provide the graded data through a data transfer or by entering the graded data on the study website. These data will remain in the study database and will not be provided to the clinical site. |
| 1310 | 9.2 Study Records Retention |
| 1311<br>1312<br>1313 | Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH E6 and regulatory and institutional requirements for the protection of confidentiality of participants. |
| 1314<br>1315<br>1316<br>1317<br>1318 | Study documents will be retained for a minimum of six (6) years from the date on which the CC receives IRB approval to close the study. These documents should be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of the sponsor. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained. |
| 1319 | 9.3 Quality Assurance and Monitoring |
| 1320<br>1321<br>1322<br>1323<br>1324<br>1325 | Designated personnel from the Coordinating Center will be responsible for maintaining quality assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is conducted and data are generated, documented and reported in compliance with the protocol, Good Clinical Practice (GCP) and the applicable regulatory requirements, as well as to ensure that the rights and wellbeing of trial participants are protected and that the reported trial data are accurate, complete, and verifiable. |
| 1326<br>1327<br>1328<br>1329<br>1330<br>1331 | A risk-based monitoring (RBM) plan will be developed and revised as needed during the study, consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations — A Risk-Based Approach to Monitoring" (August 2013). <sup>29</sup> Study conduct and monitoring will conform with 21 Code of Federal Regulations (CFR) 312. <sup>30</sup> This plan describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports. |
| 1332<br>1333<br>1334<br>1335 | The data of most importance for monitoring at the site are participant eligibility and adverse events. Therefore, the RBM plan will focus on these areas. As much as possible, remote monitoring will be performed in real-time with on-site monitoring performed to evaluate the verity and completeness of the key site data. Elements of the RBM may include: |
| 1336 | • Qualification assessment, training, and certification for sites and site personnel |
| 1337<br>1338 | <ul> <li>Oversight of Institutional Review Board (IRB) coverage and informed consent<br/>procedures</li> </ul> |

| 1339<br>1340 | <ul> <li>Central (remote) data monitoring: validation of data entry, data edits/audit trail,<br/>protocol review of entered data and edits, statistical monitoring, study closeout</li> </ul> |
|---|---|
| 1341 | <ul> <li>On-site monitoring (site visits): source data verification, site visit report</li> </ul> |
| 1342 | <ul> <li>Communications with site staff</li> </ul> |
| 1343 | <ul> <li>Patient retention and visit completion</li> </ul> |
| 1344 | <ul> <li>Quality control reports</li> </ul> |
| 1345 | <ul> <li>Management of noncompliance</li> </ul> |
| 1346 | <ul> <li>Documenting monitoring activities</li> </ul> |
| 1347 | <ul> <li>Adverse event reporting and monitoring</li> </ul> |
| 1348<br>1349<br>1350<br>1351<br>1352<br>1353 | Coordinating Center representatives or their designees may visit the study facilities at any time to maintain current and personal knowledge of the study through review of records, comparison with source documents, observation and discussion of the conduct and progress of the study. The investigational site will provide direct access to all trial-related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities. |
| 1354 | 9.4 Protocol Deviations |
| 1355<br>1356<br>1357 | A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure requirements. The noncompliance may be either on the part of the participant, the investigator, or the study site staff. |
| 1358<br>1359<br>1360<br>1361<br>1362 | A significant (or major) deviation is any deviation that departs from the established materials in such a way that it poses an increase in the risk to the study participants, adversely affects the welfare, rights, or safety of the research study participants, or negatively influences the scientific study integrity. As a result of significant deviations, corrective and preventive actions are to be developed by the site and implemented promptly. |
| 1363<br>1364 | The site PI and study staff are responsible for knowing and adhering to their IRB/EC requirements. |

#### **Chapter 10: Ethics/Protection of Human Participants** 1365 10.1 Ethical Standard 1366 The Principal Investigator (PI) will ensure that this study is conducted in full conformity with 1367 Regulations for the Protection of Human Participants of Research in accordance with ICF 1368 E6/GCP, EC requirements, and local laws and regulations, as applicable. 1369 10.2 Institutional Review Boards 1370 1371 The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the IRB for review and approval. Approval of both the protocol and the consent 1372 1373 form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All 1374 changes to the consent form will be IRB approved; a determination will be made regarding 1375 whether previously consented participants need to be re-consented. 1376 **10.3 Informed Consent Process** 1377 10.3.1 Consent Procedures and Documentation 1378 1379 Informed consent is a process that is initiated prior to the individual's agreeing to participate in 1380 the study and continues throughout the individual's study participation. Extensive discussion of risks and benefits of participation will be provided to the participants and their families. Consent 1381 forms will be IRB-approved, and the participant will be asked to read and review the document. 1382 The investigator will explain the research study to the participant and answer any questions that 1383 may arise. All participants will receive a verbal explanation in terms suited to their 1384 comprehension of the purposes, procedures, and potential risks of the study and of their rights as 1385 research participants. Participants will have the opportunity to carefully review the written 1386 consent form and ask questions prior to signing. 1387 The participants will have the opportunity to discuss the study with their surrogates or think 1388 about it prior to agreeing to participate. The participant will sign the informed consent document 1389 prior to any procedures being done specifically for the study. The participants may withdraw 1390 consent at any time throughout the course of the trial. A copy of the informed consent document 1391 will be given to the participants for their records. The rights and welfare of the participants will 1392 be protected by emphasizing to them that the quality of their medical care will not be adversely 1393 affected if they decline to participate in this study. 1394 10.3.2 Participant and Data Confidentiality 1395 Participant confidentiality is strictly held in trust by the participating investigators, their staff, 1396 1397 and the sponsor(s) and their agents. This confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. 1398 1399 Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study, or the data will be released to any 1400

The study monitor, other authorized representatives of the sponsor, representatives of the IRB, 1402 1403

unauthorized third party without prior written approval of the sponsor.

regulatory agencies or company supplying study product may inspect all documents and records

| 1404<br>1405<br>1406 | required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) for the participants in this study. The clinical study site will permit access to such records. |
|---|---|
| 1407<br>1408<br>1409<br>1410 | The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, institutional policies, or sponsor requirements. |
| 1411<br>1412<br>1413<br>1414<br>1415<br>1416<br>1417<br>1418<br>1419 | Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the FFB Consortium Coordinating Center, located at the Jaeb Center for Health Research in Tampa, FL. This will not include the participant's contact or identifying information, unless otherwise specified in the informed consent form. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by clinical sites and by the FFB Consortium Coordinating Center research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at the FFB Consortium Coordinating Center. |
| 1420 | 10.3.3 Future Use of Stored Specimens and Data |
| 1420<br>1421<br>1422<br>1423<br>1424<br>1425 | 10.3.3 Future Use of Stored Specimens and Data With the participant's approval and as approved by the IRB/ECs, de-identified biological skin fibroblasts and blood samples collected for analysis will be stored at The Kennedy Krieger Institute until the FFB Study Team notifies them in writing to destroy the samples. The blood samples will be destroyed one (1) year after the end of the study. The skin biopsy samples will be stored indefinitely with the participant's consent. |
| 1421<br>1422<br>1423<br>1424 | With the participant's approval and as approved by the IRB/ECs, de-identified biological skin fibroblasts and blood samples collected for analysis will be stored at The Kennedy Krieger Institute until the FFB Study Team notifies them in writing to destroy the samples. The blood samples will be destroyed one (1) year after the end of the study. The skin biopsy samples will |
| 1421<br>1422<br>1423<br>1424<br>1425 | With the participant's approval and as approved by the IRB/ECs, de-identified biological skin fibroblasts and blood samples collected for analysis will be stored at The Kennedy Krieger Institute until the FFB Study Team notifies them in writing to destroy the samples. The blood samples will be destroyed one (1) year after the end of the study. The skin biopsy samples will be stored indefinitely with the participant's consent. |

1436 1437 possible after the study is completed.

# **Chapter 11: References**

1439

- 1440 1. Wang T, Lawler AM, Steel G, Sipila I, Milam AH, Valle D. Mice lacking ornithinedelta-aminotransferase have paradoxical neonatal hypoornithinaemia and retinal degeneration. *Nat Genet.* 1995;11(2):185-190.
- Valle D, Simell O. The Hyperornithinemias. In: Valle DL, Antonarakis S, Ballabio A,
   Beaudet AL, Mitchell GA, eds. *The Online Metabolic and Molecular Bases of Inherited Disease*. New York, NY: McGraw-Hill Education; 2019.
- Valle D, Kaiser-Kupfer MI, Del Valle LA. Gyrate atrophy of the choroid and retina:

  deficiency of ornithine aminotransferase in transformed lymphocytes. *Proceedings of the National Academy of Sciences of the United States of America*. 1977;74(11):5159-5161.
- Mitchell GA, Brody LC, Looney J, et al. An initiator codon mutation in ornithine-deltaaminotransferase causing gyrate atrophy of the choroid and retina. *The Journal of clinical investigation*. 1988;81(2):630-633.
- Mitchell GA, Looney JE, Brody LC, et al. Human ornithine-delta-aminotransferase.
   cDNA cloning and analysis of the structural gene. *The Journal of biological chemistry*.
   1988;263(28):14288-14295.
- Mitchell GA, Brody LC, Sipila I, et al. At least two mutant alleles of ornithine deltaaminotransferase cause gyrate atrophy of the choroid and retina in Finns. *Proceedings of the National Academy of Sciences of the United States of America*. 1989;86(1):197-201.
- Honor Table 7. Brody LC, Mitchell GA, Obie C, et al. Ornithine delta-aminotransferase mutations in gyrate atrophy. Allelic heterogeneity and functional consequences. *J Biol Chem.* 1992;267(5):3302-3307.
- Michaud J, Thompson GN, Brody LC, et al. Pyridoxine-responsive gyrate atrophy of the choroid and retina: clinical and biochemical correlates of the mutation A226V. *Am J Hum Genet.* 1995;56(3):616-622.
- Lemay JF, Lambert MA, Mitchell GA, et al. Hyperammonemia-hyperornithinemiahomocitrullinuria syndrome: neurologic, ophthalmologic, and neuropsychologic examination of six patients. *J Pediatr*. 1992;121(5 Pt 1):725-730.
- 1467 10. Camacho JA, Obie C, Biery B, et al. Hyperornithinaemia-hyperammonaemia-homocitrullinuria syndrome is caused by mutations in a gene encoding a mitochondrial ornithine transporter. *Nat Genet.* 1999;22(2):151-158.
- 1470 11. Palmieri F, Scarcia P, Monné M. Diseases Caused by Mutations in Mitochondrial Carrier Genes SLC25: A Review. *Biomolecules*. 2020;10(4).
- 12. Balfoort BM, Buijs MJN, Ten Asbroek A, et al. A review of treatment modalities in gyrate atrophy of the choroid and retina (GACR). *Mol Genet Metab.* 2021;134(1-2):96-116.
- Valle D, Walser M, Brusilow S, Kaiser-Kupfer MI, Takki K. Gyrate atrophy of the choroid and retina. Biochemical considerations and experience with an arginine-restricted diet. *Ophthalmology*. 1981;88(4):325-330.
- 1478 14. Kaiser-Kupfer MI, de Monasterio F, Valle D, Walser M, Brusilow S. Visual results of a long-term trial of a low-arginine diet in gyrate atrophy of choroid and retina.

  Ophthalmology. 1981;88(4):307-310.

- Valle D, Walser M, Brusilow SW, Kaiser-Kupfer M. Gyrate atrophy of the choroid and retina: amino acid metabolism and correction of hyperornithinemia with an arginine-deficient diet. *J Clin Invest.* 1980;65(2):371-378.
- 1484 16. Kaiser-Kupfer MI, de Monasterio FM, Valle D, Walser M, Brusilow S. Gyrate atrophy of 1485 the choroid and retina: improved visual function following reduction of plasma ornithine 1486 by diet. *Science*. 1980;210(4474):1128-1131.
- 1487 17. Kaiser-Kupfer MI, Caruso RC, Valle D, Reed GF. Use of an arginine-restricted diet to slow progression of visual loss in patients with gyrate atrophy. *Arch Ophthalmol*. 2004;122(7):982-984.
- 1490 18. Kaiser-Kupfer MI, Caruso RC, Valle D. Gyrate atrophy of the choroid and retina. Long-1491 term reduction of ornithine slows retinal degeneration. *Arch Ophthalmol*. 1492 1991;109(11):1539-1548.
- 1493 19. Wang T, Milam AH, Steel G, Valle D. A mouse model of gyrate atrophy of the choroid and retina. Early retinal pigment epithelium damage and progressive retinal degeneration.

  1494 *J Clin Invest.* 1996;97(12):2753-2762.
- Wang T, Steel G, Milam AH, Valle D. Correction of ornithine accumulation prevents retinal degeneration in a mouse model of gyrate atrophy of the choroid and retina.

  Proceedings of the National Academy of Sciences of the United States of America.

  2000;97(3):1224-1229.
- Sipilä I, Simell O, Arjomaa P. Gyrate atrophy of the choroid and retina with hyperornithinemia. Deficient formation of guanidinoacetic acid from arginine. *J Clin Invest.* 1980;66(4):684-687.
- Vannas-Sulonen K, Sipilä I, Vannas A, Simell O, Rapola J. Gyrate atrophy of the choroid and retina. A five-year follow-up of creatine supplementation. *Ophthalmology*. 1985;92(12):1719-1727.
- Heinänen K, Näntö-Salonen K, Komu M, et al. Creatine corrects muscle 31P spectrum in gyrate atrophy with hyperornithinaemia. *Eur J Clin Invest*. 1999;29(12):1060-1065.
- Hanna-El-Daher L, Braissant O. Creatine synthesis and exchanges between brain cells:
  What can be learned from human creatine deficiencies and various experimental models?

  Amino Acids. 2016;48(8):1877-1895.
- Du J, Zhu S, Lim RR, Chao JR. Proline metabolism and transport in retinal health and disease. *Amino Acids*. 2021;53(12):1789-1806.
- Elnahry AG, Elnahry GA. Gyrate Atrophy of the Choroid and Retina: A Review. *European Journal of Ophthalmology.* 2021:11206721211067333.
- Food and Drug Administration. Rare Diseases: Natural History Studies for Drug Development. In. *Draft Guidance for Industry*, 2019.
- 1517 28. Ying GS, Maguire MG, Glynn RJ, Rosner B. Tutorial on Biostatistics: Longitudinal
  1518 Analysis of Correlated Continuous Eye Data. *Ophthalmic epidemiology*. 2021;28(1):31519 20.
- Food and Drug Administration. Guidance for Industry Oversight of Clinical Investigations A Risk-Based Approach to Monitoring. In:2013.
- 1522 30. Food and Drug Administration. 21 Code of Federal Regulations (CFR) 312. In:2022.